

# NON-INTERVENTIONAL STATISTICAL ANALYSIS PLAN FOR SECONDARY DATA COLLECTION STUDY

# **VERSION HISTORY**

| pose of changes is to further clarify and resent data. The vast majority of those are made related to appendix 4 of ells. The changes do not impact data or result generation. |
|---|
| Change "main cohort" to "main study" Change "prospective Cohort" or "prospective study" to "prospective cohort study" Change "Prevan13" to "13vPnC" Change "PCV13" to "13vPnC" Change "PCV13" to "13vPnC" Appendix 1 and 2: The Table shell (Appendix 4): Add tables 4.1.2, 4.1.5, 4.2.2, 4.2.5, 5.1.2, 5.1.5, 5.2.2, 5.2.5, and change the serial number for other tables accordingly (eg, 4.1.2 to 4.1.3) − (Note: these tables were developed and included in the SAP version 1.0 but were left out accidentally at the time to attach them in the Table Shell, Appendix 4). Add variable "Febrile seizures" for tables 2.1, 4.1.1-4.2.6 Drop variable "Highest temperature for each day fever is reported" for tables 5.1.1-5.2.6 Add variable "Residential area" for table 1.1, 1.2, 3.1, 3.2 Change "children" to "participants" Change "subjects" to "participants" Change "Safety Outcomes" to "Safety Outcomes of Interest" Format "0<-2" as "0- ≤2", "2<-4" as "2- ≤4", etc. |

| administration" |
|------------------------------------------------------------------------|
| o Change "Seizures (including febrile |
| seizures)" to "All Seizures" |
| o Change "Seizures (NOT including febrile seizures)" to "All Seizures" |
| o Other format changes include to |
| change n to n (%) in the row titles, or |
| drop n (%) in the column titles, and |
| refine some footnotes. |



# **Non-Interventional Study Protocol**

B1851193

# An observational safety study for Prevenar 13 among Chinese children

# Statistical Analysis Plan (SAP)

Version: <2.0>

Author: PPD , Global Medical Epidemiology, Worldwide Medical & Safety, Worldwide Research, Development & Medicine, Pfizer Inc, New York, NY 10017, USA

Date: 07 Januray 2021

# TABLE OF CONTENTS

| LIST OF TABLES | 4 |
|-----------------------------------------------------|------|
| LIST OF FIGURES | 5 |
| APPENDICES | 5 |
| 1. AMENDMENTS FROM PREVIOUS VERSION(S) | 6 |
| 2. INTRODUCTION | 6 |
| 2.1. Study Objectives | 7 |
| 2.2. Study DESIGN | 8 |
| 2.2.1. Study population | 8 |
| 2.2.2. Data Source | 9 |
| 2.2.3. Yinzhou EHR Database | 9 |
| 3. HYPOTHESES AND DECISION RULES | 11 |
| 4. ANALYSIS SETS/POPULATIONS | 11 |
| 4.1. Analysis Set | 11 |
| 4.1.1. Inclusion Criteria | 11 |
| 4.1.2. Exclusion Criteria | 11 |
| 4.2. Sub analysis set | 11 |
| 4.3. Subgroups | 11 |
| 5. ENDPOINTS AND COVARIATES | 12 |
| 5.1. Safety Endpoints | 12 |
| 5.2. Covariates | 12 |
| 6. HANDLING OF MISSING VALUES | 14 |
| 7. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | S 14 |
| 7.1. Descriptive Analysis | 14 |
| 7.2. Validation of ICD Codes | 16 |
| 7.3. Summary of Analyses | 17 |
| 8. LIST OF TABLES AND TABLE SHELLS | |
| 9. REFERENCES | |
| 10. APPENDICES | 20 |
| LIST OF TABLES | |
| Table 1. Variables and Roles | 12 |

# LIST OF FIGURES

| Figure 1. | Flow Chart of Study Period | 8 |
|-----------|-------------------------------------|----|
| Figure 2. | Flow Chart for Study Populations | 9 |
| Figure 3. | Procedures for the Validation Study | 17 |
| | APPENDICES | |

Appendix 3. Other vaccines potentially administrated on the same date with

## 1. AMENDMENTS FROM PREVIOUS VERSION(S)

None.

#### 2. INTRODUCTION

Pneumococcal disease is a leading cause of serious illness throughout the world.<sup>1</sup> It is an infection caused by Streptococcus pneumoniae bacteria ("pneumococcus"). These bacteria can result in both invasive diseases such as bacteremic pneumonia, septicemia, and meningitis, and non-invasive diseases, such as pneumonia, otitis media, and sinus infections. One of the key risk factors of pneumococcal diseases is age, with children younger than 2 years of age and the elderly being at the highest risk of developing pneumococcal-related infection.<sup>1</sup> Pneumococcal disease is estimated to be the leading cause of vaccine-preventable morbidity and mortality among children younger than 5 years both globally and in China.<sup>1</sup> At least 1 million children die of pneumococcal disease every year, most of these being young children in developing countries.<sup>2</sup> In China alone, approximately 30 thousand children in this age group die due to pneumococcal disease every year.<sup>3</sup>

Currently, several approved vaccines to prevent S. pneumoniae infections are available on the market, including the 10-, and 13-valent pneumococcal conjugate vaccines (10 vPnC; Synflorix, GlaxoSmithKline and 13vPnC; Prevnar 13, Pfizer, respectively), and the 23-valent pneumococcal polysaccharide vaccine (PPSV23; Pneumovax, SanofiPasteurMSD [in the US, Merck]). 13vPnC was approved in the European Union in December 2009 for the prevention of Invasive Pneumococcal Disease (IPD), pneumonia and acute otitis media caused by S. pneumoniae in infants, children and adolescents from 6 weeks to 17 years of age, and in the United States in February 2010 for the prevention of IPD and otitis media caused by S. pneumoniae in children 6 weeks through 5 years of age.

13vPnC is in use in the national childhood immunization programs in many countries and contains polysaccharides from the 7 serotypes included in the original 7vPnC (4, 6B, 9V, 14, 18C, 19F, and 23F) and an additional 6 serotypes (1, 3, 5, 6A, 7F, and 19A), all conjugated to cross-reactive material 197. It has been shown that the 6 additional serotypes in 13vPnC increase coverage for IPD prevention in children <5 years of age from 74% to 88% globally. Importantly, the additional serotypes in 13vPnC are associated with a high percentage of pneumococcal disease in the developing world. 5,6

In October 2016, 13vPnC was approved in China for the prevention of invasive disease (including bacteremic pneumonia, meningitis, septicemia, and bacteremia) caused by Streptococcus pneumoniae for infants and children aged 6 weeks to 15 months. 13vPnC is recommended as a series of four doses, one dose at each of these ages: 2 months; 4 months; 6 months; 12 through 15 months. Vaccines in China are classified into two categories. Type I vaccines are mandatory and provided for citizens by the government free of charge, and infants and children should get immunized according to the government's regulations. These vaccines include tuberculosis (Bacillus Calmette—Guérin), diphtheria/tetanus/ pertussis, oral polio, measles/mumps/rubella, hepatitis B, hepatitis A, meningococcal, and Japanese encephalitis. Type II vaccines are ones

available on the private market for use on a voluntary base at the purchaser's expense. They consist of Haemophilus influenzae type b (Hib), pneumococcal conjugate, rotavirus (RV), inactivated polio (IPV), varicella, human papillomavirus, and influenza vaccines. In China, all type I and type II vaccines are administrated at China Centers for Disease Control and Prevention (CDC) immunization clinics.

13vPnC has a favorable benefit-risk profile. Based on data from clinical trials and the worldwide safety experiences after authorization, convulsions/seizures, fever, apnea, and anaphylaxis/hypersensitivity are identified as known or potential risks associated with 13vPnC among young children.<sup>7,8</sup>

To monitor these known and potential risks for 13vPnC among Chinese children receiving 13vPnC in China, an observational study using a population-based electronic health record (EHR) database from May 1<sup>st</sup>, 2017 to July 31<sup>st</sup>, 2020 in Yinzhou district of Ningbo city in China will be conducted in a real world setting. Yinzhou is one of the largest districts in economically developed Ningbo city. Children exposed to 13vPnC in Yinzhou district are representative of those children likely receiving 13vPnC in China given that only families with sufficient financial resources can afford 13vPnC. In addition, the coverage for 7vPnC in Yinzhou district was similar to that in the published literature in China.<sup>9</sup> As a population-based database, Yinzhou EHR database consists of complete immunization records and healthcare data of all children in the district. This allows for the possibility of monitoring the safety of 13vPnC in the context of routine medical care from outpatient visits to inpatient care and provides greater generalizable findings.

This observational safety study is a post authorization commitment (PAC) to fulfill the key monitoring activity requirement of the National Medical Products Administration (NMPA) in China.

# 2.1. Study Objectives

The overall objective of this observational study is to expand the understanding of the safety profile of 13vPnC in Chinese pediatric populations.

Specific objectives of the study are to:

- Estimate incidence rates (per 1,000 person-days at risk and per 1,000 doses) of safety outcomes of interest (SOIs) including seizures (including febrile seizures), urticaria and angioedema, apnea, and fever for the periods of 0 through 3 days (with 0 indicating the day of vaccination), 4 through 7 days, and 0 through 7 days after the 13vPnC vaccination by all doses and by each dose in the main study based on Yinzhou EHR database between 1 May 2017 and 31 July 2020.
- Estimate the incidence rates (per 1,000 person-days at risk and per 1,000 doses) of the SOIs above after the 13vPnC vaccination by all doses and by each dose in a sub-population of the main study through a prospective cohort study between 1 August 2018 and 31 July 2020.

All SOIs are acute events and are likely to occur within 7 days post-vaccination based on the known safety profile of 13vPnC as well as biologic plausibility of these events occurring after vaccination.<sup>7,8</sup>

# 2.2. Study DESIGN

This is an observational study based on a population-based EHR database. In addition, a validation study including validation of ICD-10 codes or ICD-10 code based algorithm for identifying all SOIs and a prospective cohort study in a sub-population of the main study will be conducted in order to offset the potential biased results from the main study because of potential misclassification of the SOIs due to miscoding and/or undercoding of ICD-10 codes used to identify these safety outcomes in the EHR database.

Figure 1. Flow Chart of Study Period



Note: The end of enrolment for both Prospective Cohort Study as well as the main study is the same-July 24, 2020 although we don't actively enroll patients in the main study. In other words, any doses received after July 24, 2020 won't be included. For both studies, we allow a 7-day follow up period for each dose. Thus, the study end date for both studies is July 31, 2020.

#### 2.2.1. Study population

The main study population consists of eligible children aged 1-24 months receiving at least one dose of 13vPnC recorded in Yinzhou EHR database between 1 May 2017 and 24 July 2020 (i.e. one week prior to the end of the study) (Figure 2).



Figure 2. Flow Chart for Study Populations

#### 2.2.2. Data Source

Since 2014, via collaboration with academic institutions in China, Pfizer has been evaluating various observational data sources in China and has determined that they provide potential value to post-marketing drug safety studies, particularly population-based EHRs. Yinzhou EHR database is selected for this study because this population-based EHR database consists of complete immunization records and healthcare data of all children in the district.

# 2.2.3. Yinzhou EHR Database

Yinzhou is one of the largest districts of economically developed Ningbo city in Zhejiang province, China and consists of approximately 1.6 million populations (740,000 permanent residents and 860,000 temporary residents). The Yinzhou EHRs include data from three main sources (Figure 3):

• Yinzhou CDC databases;

- Healthcare data including EMRs, claims and e-prescriptions from hospitals and community health centers within the district;
- Healthcare data including EMRs, claims and e-prescriptions from the Women and Children's hospital of Ningbo city.

Figure 3. Components of Yinzhou EHR Database



Data from these data sources are entered into Yinzhou EHR database in real time. These data sources are linked via each child's unique personal identification number (termed the national identification (NID) number) used by each resident throughout life in China. In a situation where children do not yet have a NID number, data of those children are matched by names of children, dates of birth, names of parents/legal guardians, or home addresses.

- a. **Yinzhou CDC database:** There are two CDC databases (ie, Immunization Administration Registry and CDC AEFIS) in the district. The Immunization Administration Registry includes immunization data at CDC immunization clinics for both type I and type II vaccines for all children aged <7 years. The AEFIS is a passive surveillance system and collects AEFIs reports. All cases reported to AEFIS are to be investigated, with the exception of common adverse reactions that have a clear diagnosis (eg, fever, redness, and swelling on the injection site; induration).
- b. **Healthcare data from hospitals and community health centers within the district:** Yinzhou district collect healthcare data of its residents from hospitals (3 tertiary general hospitals and 1 specialized hospital) and community health centers (20) within the district including inpatient and outpatient visits from all hospitals and outpatient visits from all community health centers within the district.

c. Healthcare data from the Women and Children's Hospital of Ningbo city:

The Women and Children's Hospital of Ningbo city is the only children hospital in the city. It is essential to have data from this hospital being part of Yinzhou EHR database because this hospital is very likely to be the hospital of choice if families would seek medical care for their children outside hospitals of Yinzhou district.

#### 3. HYPOTHESES AND DECISION RULES

NA: This is a descriptive study

#### 4. ANALYSIS SETS/POPULATIONS

An overall analysis population is defined in Figure 2, Section 2.2.

# 4.1. Analysis Set

#### 4.1.1. Inclusion Criteria

Children must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- For main study, all children must be aged 1 to 24 months and receive at least one dose of 13vPnC between 1 May 2017 and 24 July 2020 where the first dose is received before or on 24 July 2020 since a 7-day post-vaccination follow-up for each dose in each child receiving 13vPnC is needed.
- The index date for this overall cohort of the main study is defined as the 1<sup>st</sup> date that an eligible child receives any dose of 13vPnC in the series between 1 May 2017 and 24 July 2020.

#### 4.1.2. Exclusion Criteria

There are no exclusion criteria for this study.

#### 4.2. Sub analysis set

For the prospective cohort study in a sub-population of the main study, eligible children must receive the first dose of 13vPnC between 1 August 2018 and 24 July 2020 and an informed consent must be obtained from parents/legal guardians (Figure 2).

• The index date for this prospective cohort study as a sub set of the main study is defined as the 1<sup>st</sup> date that an eligible child receives the 1<sup>st</sup> dose of 13vPnC in the series between 1 August 2018 and 24 July 2020

#### 4.3. Subgroups

Subgroup analysis may be considered, including but not limited to subgroup analyses by age, dosage, and follow-up length.

#### 5. ENDPOINTS AND COVARIATES

Five safety outcomes will be evaluated in this study. ICD 10 codes and risk windows for these outcomes are described in details in section 5.1. As we are evaluating acute events after each dose among children aged 1-24 months, the risk windows are very short. The baseline period varies by each child and is defined as the period between the date entering the study (i.e. the enrolment data in the study dataset) and the 1<sup>st</sup> date receiving any available dose at age 1-24 months (main study). Demographic characteristics at time entering the study and age at the time receiving each dose of 13vPnC will be described (see Section 7)

## 5.1. Safety Endpoints

| Outcome* | Main Study | Porspective Cohort | Risk window for each dose and for all doses |
|---|---|---|---|
| Seizures (including febrile seizures) | Appendix 1 (ICD 10 code list for the Outcome of Interests) | | 0-3 days, 4-7 days, 0-7 days |
| Seizures (NOT including febrile seizures) | | Reported Terms | 0-3 days, 4-7 days, 0-7 days |
| Febrile seizures | | Reported Terms | 0-3 days, 4-7 days, 0-7 days |
| Urticaria and angioedema | Appendix 1(ICD 10 code list for the Outcome of Interests) | Reported Terms | 0-3 days, 4-7 days, 0-7 days |
| Apnea | Appendix 1 (ICD 10 code list for the Outcome of Interests) | Reported Terms | 0-3 days, 4-7 days, 0-7 days |
| Fever | Appendix 1 (ICD 10 code list for the Outcome of Interests) | Reported Terms (≥38°C) | 0-3 days, 4-7 days, 0-7 days |
| Highest<br>temperature for<br>each day fever | | Reported Terms | 0-3 days, 4-7 days, 0-7 days |

<sup>\*</sup>Please note, ICD codes will be used to capture these events for the main study but reports of these events from parents will be used for the prospective cohort study.

#### 5.2. Covariates

**Table 1.** Variables and Roles

| Variable | Role | Operational definition |
|---|---|---|
| Age | Demographic | Age at index date, age at entering into study, age at 1 <sup>st</sup> diagnosis depending on the reporting purposes (see Table shell – Appendix 4) |
| Gender | Demographic | Female, Male |
| Residency Status | Demographic | Permanent residents, Temporal |

| | | residents at time entering the study |
|---|---|---|
| Known allergies | Medical history | Only in prospective cohort study, reported during the 1 <sup>st</sup> visit (Yes/No) |
| Gestational Age | Medical history | Full term (>=37 weeks), Preterm (<37 weeks) reported during the 1st visit in prospective cohor; or diagnosis codes prior to the 1st date of a dose available in the database |
| Birth weight | Medical history | Normal (>=2500 g), Low birth weight (<2500 g) reported during the 1 <sup>st</sup> visit in prospective cohort study; or diagnosis codes prior to the 1 <sup>st</sup> date of a dose available in the database |
| Sickle cell disease | Medical history | In prospective cohort study, reported during the 1 <sup>st</sup> visit (Yes/No) In main study, look at the diagnosis codes prior to the 1 <sup>st</sup> date of a dose available in the database (Appendix 2– ICD 10 code list for the covarites) |
| History of febrile seizure | Medical history | In prospective cohort study, reported during the 1 <sup>st</sup> visit (Yes/No) In main study, look at the diagnosis codes prior to the 1 <sup>st</sup> date of a dose available in the database (Appendix 1) |
| History of other seizures | Medical history | In prospective cohort study, reported during the 1 <sup>st</sup> visit (Yes/No) In main study, look at the diagnosis codes prior to the 1 <sup>st</sup> date of a dose available in the database (Appendix 2- ICD 10 code list for the covarites) |
| History of urticaria | Medical history | In prospective cohort study, reported during the 1 <sup>st</sup> visit (Yes/No) In main study, look at the diagnosis codes prior to the 1 <sup>st</sup> date of a dose available in the database (Appendix 2- ICD 10 code list for the covarites) |
| History of angioedema | Medical history | In prospective cohort study, reported during the 1 <sup>st</sup> visit (Yes/No) In main study, look at the diagnosis codes prior to the 1 <sup>st</sup> date of a dose available in the database (Appendix 2- ICD 10 |

| | | code list for the covarites) |
|---|---|---|
| History of apnea | Medical history | In prospective cohort study, reported during the 1 <sup>st</sup> visit (Yes/No) In main study, look at the |
| | | diagnosis codes prior to the 1 <sup>st</sup> date of a dose available in the database (Appendix 1) |
| Fever at the date prior to 13vPnC vaccination | Medical history | In prospective cohort study, reported during the 1 <sup>st</sup> visit (Yes/No) In main study, look at the diagnosis codes prior to the 1 <sup>st</sup> date of a dose available in the database (Appendix 1) |
| Smoking in the family | Covariate | Only in prospective cohort study, reported during the 1 <sup>st</sup> visit (Yes/No) |
| Season of diagnosis for each safety outcome of interest | Covariate | Date of diagnosis of outcome of interests |
| Hospitalization for each safety outcome of interest | Covariate | Admission to hospital for the outcome of the interests: 1). In prospective cohort study, (Yes/No), reported during each visit) 2). In main study, using admission or discharge diagnosis to be the outcome of interests |
| Use of antipyretics post-vaccination | Covariate | Only in prospective cohort study, (Yes/No), reported during each visit) |
| Date of each dose of 13vPnC vaccination (based on barcode scanning) | Exposure | Date of administration |
| Other vaccines administrated the same date with 13vPnC | Co-administration | Date of administration (Appendix 3- Other vaccines potentially administrated on the same date with 13vPnC) |

# 6. HANDLING OF MISSING VALUES

No imputation for missing values will be performed.

# 7. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

### 7.1. Descriptive Analysis

Means, medians, and standard deviations will be provided for continuous variables. Numbers and percentages will be provided for dichotomous variables or categorical variables. Frequency distributions of age at the time receiving each dose of 13vPnC, gender, residential status, birthweight, gestational age, year of 13vPnC vaccinations, co-administration of other vaccines at the same date, and medical history will be described (Appendix 4: Table shell). In addition, frequency distributions of the number of SOIs by age, gender, residential status, season of vaccination, hospitalization, and year of 13vPnC

vaccinations will also be described (Appendix 4: Table shell). The frequency distributions mentioned above will be tabulated for both the main study and the prospective cohort study in the sub-population of the main study.

The incidence rate and its 95% CI for each safety outcome will be calculated per 1,000 person-days at risk and per 1,000 doses. For the former, the incidence rate will be calculated as the number of children exposed to each dose who experience the event during the specified risk window (ie, 0-3 days, 4-7 days, and 0-7 days post-vaccination) divided by the observed time at risk, multiply by 1000 (i.e. IR per 1000 person-days at risk). For the latter, the incidence rate will be calculated as the number of children exposed to each dose who experience the event during the specified risk window (ie, 0-3 days, 4-7 days, and 0-7 days post-vaccination) divided by the number of child receiving this specific dose, multiply by 1000 (ie. IR per 1000 doses). The incidence rate for each safety outcome will also be stratified by potential risk factors such as age group, gender, residence status, co-adminstration of other vaccines on the same date, season of adminstration of 13vPnC (Appendix 4: Table shell). The incidence rates will be estimated for both the main study and the prospective cohort study in the sub-population of the main study.

#### 7.2. Validation of ICD Codes

To evaluate the accuracy of the ICD-10 codes or ICD-10 codes based algorithm for identifying all SOIs in the main study, relevant medical records of children having the ICD codes for these events are going to be obtained from hospitals within Yinzhou district and Women and Children's hospital of Ningbo city and outpatient medical records from community health centers within the district by Yinzhou CDC. A data abstraction form will be used to abstract data from the medical records. The abstracted data will be sent to an adjudication committee to determine whether the identified potential case is a true case. Then the adjudicated outcomes will be entered into the validation study database for analyses. The procedures for the validation study is described in Figure 3. The following analyses of positive predicted value (PPV), sensitivity (SE), specificity (SP), positive percent of agreement (PPA), and negative percent of agreement (NPA) will be calculated for main study and prospective cohort study respective performed (Appendix 4: Table shell).

The PPV of an ICD-10 code or ICD-10 code based algorithm used to identify the SOIs against adjudicated outcomes based on medical records as a gold standard will be calculated for the validation of these codes in the main study.

- The PPV of a reported safety outcome of interest by parents/legal guardians that requires medical attentions against the adjudicated safety outcome based on medical records of children as a gold standard will be calculated in the prospective cohort study in the sub-population of the main study.
- Among children who participate in both the main study and the prospective cohort study, sensitivity and specificity of an ICD code or ICD-10 code based algorithm identifying seizures or apnea in the main study will be calculated using the adjudicated safety outcome in the prospective cohort study as a reference standard (ie, a gold standard).

• A positive percent of agreement and a negative percent of agreement will be estimated between an ICD code or ICD-10 code based algorithm identifying fever or urticaria and angioedema in the main study and the reported fever or urticaria and angioedema by parents/legal guardians in the prospective cohort study as a non-reference standard (ie, a non-gold standard).

Validation Study Validation of ICD codes Prospective cohort study in a used to identify safety sub-population outcomes of interest Recruitment of parents/legal Abstract data from medical charts professionals at CDC If child receives immunization clinics medial care for afety outcomes of interest Abstracted data Parents/legal guardians reviewed by complete paper or online adjudication committee initial and follow-up questionnaires via phone or face-to-face interviews Adjudication outcomes Completed questionnaires Validation study database Linked via national ID or other identifiable data Main study database based

Figure 3. Procedures for the Validation Study

All data analysis will be executed using statistical software SAS version 9.4 or later.

on Yinzhou EHR database

# 7.3. Summary of Analyses

| | Analysis Set | Supports<br>Protocol<br>Objective<br>Number | Subgroup | Statistical<br>Method | Covariates/Strata | Missing<br>Data |
|---|---|---|---|---|---|---|
| Characteristics of children | All enrolled children | 1 and 2 | NA | Descriptive analysis | NA | Included |
| Incidence rate | All enrolled children | 1 and 2 | Dose, age,<br>gender,<br>residence<br>status,<br>season, co-<br>committant<br>drugs | Descriptive<br>analysis | Stratified by the subgroups | Excluded |
| ICD code<br>validation | All cases<br>where<br>medical<br>charts or data<br>on medical<br>charts are<br>available | 1 and 2 | NA | PPV, SE, SP,<br>PPA, NPA* | NA | Excluded |

<sup>\*</sup>Positive predicted value (PPV), sensitivity (SE), specificity (SP), positive percent of agreement (PPA), and negative percent of agreement (NPA)

#### 8. LIST OF TABLES AND TABLE SHELLS

See Appendix 4.

#### 9. REFERENCES

- 1. WHO Centers for Disease Control and Prevention. Pneumococcal disease. In: Atkinson W, Wolfe S, Hamborsky J, eds. Epidemiology and Prevention of Vaccine-Preventable Diseases. 12th ed. Washington, DC: Public Health Foundation; 2011:233-248. Available at: http://www.cdc.gov/vaccines/pubs/pinkbook/pneumo.html.
- 2. Pneumococcal vaccines: WHO position paper. Weekly Epidemiological Record, 1999,74:177–183
- 3. O'Brien KL, et al. Burden of disease caused by Streptococcus pneumoniae in children younger than 5 years: global estimates. Lancet. 2009; 374(9693): 893-902.
- 4. Johnson HL, Deloria-Knoll M, et al. Systematic evaluation of serotypes causing invasive pneumococcal disease among children under five: the pneumococcal global serotype project. PLoS Medicine/Public Library of Science 2010;7(10).
- 5. Dinleyici EC, Yargic ZA. Current knowledge regarding the investigational 13-valent pneumococcal conjugate vaccine. Expert Rev Vaccines. 2009;8:977-986.
- 6. Hausdorff WP. The roles of pneumococcal serotypes 1 and 5 in paediatric invasive disease. Vaccine. 2007;25:2406-2412.
- 7. 13vPnC Risk Management Plan dated December 11th, 2017
- 8. Rowhani-Rahbar A, Klein NP, Dekker CL, et al. Biologically plausible and evidence-based risk intervals in immunization safety research. Vaccine 2012;31:271-7
- 9. Wagner AL, Sun X, Montgomery JP, Huang Z, Boulton ML. The impact of residency and urbanicity on Haemophilus influenzae Type b and pneumococcal immunization in Shanghai Children: a Retrospective Cohort Study. PLoS One. 2014 May 14;9(5).
- 10. Yang Y, Zhou X, Gao S, et al. Evaluation of Electronic Healthcare Databases for Post-Marketing Drug Safety Surveillance and Pharmacoepidemiology in China. Drug Safety. 2017 Aug 16.
- 11. Duffy J, Weintraub E, Hambidge S et al, Febrile Seizure Risk After Vaccination in Children 6 to 23 Months, PEDIATRICS, Volume 138, number 1, July 2018.
- 12. Tse A, Tseng HF, Greene S. K et al. Signal identification and evaluation for risk of febrile seizures in children following trivalent inactivated influenza vaccine in the Vaccine Safety Datalink Project, 2010–2011, Vaccine 30 (2012) 2024–2031.

13. Yih W. K, Kulldorff M, Sandhu S. K et al Prospective influenza vaccine safety surveillance using fresh data in the Sentinel System, Pharmacoepidemiology and Drug Safety 2016; 25: 481–492.
















# Appendix 3. Other vaccines potentially administrated on the same date with 13vPnC - highlighted in the Table 1 and Table 2 Table 1. Immunization schedule for Type I vaccines for children aged 0-2 years in China

| Age/Vaccine | Bacillus<br>Camette-<br>Guerin | Hepatitis B | Polio | Diaphtheria/pertussis<br>/Tetanus | Measles/<br>Mumps/<br>Rubella | Japanese<br>Encephalitis | Meningococcal | Hepatitis A |
|---|---|---|---|---|---|---|---|---|
| Birth | B.C.G | HBV1 | | | | | | |
| 1Month | | HBV2 | | | | | | |
| 2Months | | | OPV1 | | | | | |
| 3Months | | | OPV2 | DPT1 | | | | |
| 4Months | | | OPV3 | DPT2 | | | | |
| 5Months | | | | DPT3 | | | | |
| 6Months | | HBV3 | | | | | | |
| 6-18Months | | | | | | JEV 2dose | | |
| 8Months | | | | | MMR | | | |
| 10-22Months | | | | | | | MCV 2dose | |
| 1-2 years | | | Booster | Booster | | Booster | | HAV1 |

Table 2. Immunization schedule for Type II vaccines for children aged 0-2 years in China

| Age/Vaccines | Haemophilus<br>Influenzae<br>type b | Varicella | Rotavirus | Influenza | Pneumococca 1 | Pentaxim | IVP |
|---|---|---|---|---|---|---|---|
| Birth | | | | | | | |
| 1Month | | | | | | | |
| 2Months | Hib1 | | RV1 | | 13vPnC-1 | Pentaxim1 | IPV1 |
| 3Months | Hib2 | | RV2 | | | Pentaxim2 | IPV2 |
| 4Months | Hib3 | | RV3 | | 13vPnC-2 | Pentaxim3 | IPV3 |
| 5Months | | | | | | | |
| 6Months | | | | | 13vPnC-3 | | |
| 12-15 Months | | | | | PCV Booster | | |
| 10-22Months | Hib Booster | Varicella1 | | | | | |
| 1-2 years | | | | Influenza | Booster | Booster | Booster |

# Appendix 4. Table Shell

**Summary-TOC** 

- Table 1.1 Participant Demographics and Clinical Characteristics at Baseline Main Study
- **Table 1.2 Participant Demographics and Clinical Characteristics at Baseline Prospective Cohort Study**
- Table 2.1 Administration of 13vPnC by Dose Main Study
- Table 2.2 Administration of 13vPnC by Dose Prospective Cohort Study
- Table 3.1 Distribution of Safety Outcomes of Interest Main Study
- Table 3.2 Distribution of Safety Outcomes of Interest Prospective Cohort Study
- Table 4.1.1 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Main Study (All Age: 0-24 months)
- Table 4.1.2 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Main study (Age Stratification)
- Table 4.1.3 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Main Study (by Gender)
- Table 4.1.4 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Main Study (by Residence Status)
- Table 4.1.5 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Main study (by Co-administration of other vaccines on the same date)
- Table 4.1.6 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Main Study (by Season of administration of 13vPnC)
- Table 4.2.1 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Main Study (All Age: 0-24 months)
- Table 4.2.2 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Main study (Age Stratification)
- Table 4.2.3 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Main Study (by Gender)
- Table 4.2.4 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Main Study (by Residence Status)

- Table 4.2.5 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Main study (by Co-administration of other vaccines on the same date)
- Table 4.2.6 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Main Study (by Season of administration of 13vPnC)
- Table 5.1.1 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Prospective Cohort Study (All Age: 0-24 months)
- Table 5.1.2 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Prospective cohort study (Age Stratification)
- Table 5.1.3 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Prospective Cohort Study (by Gender)
- Table 5.1.4 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Prospective Cohort Study (by Residence Status)
- Table 5.1.5 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Prospective cohort study (by Co-administration of other vaccines on the same date)
- Table 5.1.6 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest Prospective Cohort Study (by Season of administration of 13vPnC)
- Table 5.2.1 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Prospective Cohort Study (All Age: 0-24 months)
- Table 5.2.2 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Prospective cohort study (Age Stratification)
- Table 5.2.3 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Prospective Cohort Study (by Gender)
- Table 5.2.4 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Prospective Cohort Study (by Residence Status)
- Table 5.2.5 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Prospective cohort study (by Co-administration of other vaccines on the same date)
- Table 5.2.6 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest Prospective Cohort Study (by Season of administration of 13vPnC)
- Table 6 Validation of ICD code using adjudicated safety outcome based on medical records of children as gold standard: Positive Predictive Value (PPV)
- Table 6.1.1 Validation of ICD code (Main Study): Seizures (including febrile seizures)
- Table 6.1.2 Validation of ICD code (Main Study): Urticaria and angioedema

- Table 6.1.3 Validation of ICD code (Main Study): Apnea
- Table 6.1.4 Validation of ICD code (Main Study): Fever
- Table 6.2.1 Validation of ICD code (Prospective Cohort Study): Seizures (including febrile seizures)
- Table 6.2.2 Validation of ICD code (Prospective Cohort Study): Urticaria and angioedema
- Table 6.2.3 Validation of ICD code (Prospective Cohort Study): Apnea
- Table 6.2.4 Validation of ICD code (Prospective Cohort Study): Fever
- Table 7 Validation of ICD code using adjudicated safety outcome in the Prospective Cohort Study as a reference standard: Sensitivity and Specificity
- Table 7.1.1 Validation of ICD code using adjudicated safety outcome in the Prospective Cohort Study as a reference standard: Seizures (including febrile seizures)
- Table 7.1.2 Validation of ICD code using adjudicated safety outcome in the Prospective Cohort Study as a reference standard: Apnea
- Table 8 Validation of ICD code using the reported terms by parents/legal guardians in the Prospective Cohort Study as a non-reference standard: Positive Percentage Agreement (PPA) and Negative Percentage Agreement (NPA)
- Table 8.1.1 Validation of ICD code using the reported terms by parents/legal guardians in the Prospective Cohort Study as a non-reference standard: Urticaria and angioedema
- Table 8.1.2 Validation of ICD code using the reported terms by parents/legal guardians in the Prospective Cohort Study as a non-reference standard: Fever

| | Overall<br>n (%) |
|------------------------------------------|------------------|
| | XXX |
| Number of Participants | AAA |
| Age at entering the study [month] | XXX (XX.X) |
| Mean (SD) | |
| Median | XXX |
| Minimum | XXX |
| Maximum | XXX |
| Age groups at entering the study (month) | |
| 0- ≤2 | XXX |
| 2-≤4 | XXX |
| 4- ≤6 | XXX |
| 6- ≤8 | XXX |
| 8- ≤10 | XXX |
| 10- ≤12 | XXX |
| 12- ≤14 | XXX |
| 14- ≤16 | XXX |
| 16-≤18 | XXX |
| 18- ≤20 | XXX |
| 20- ≤22 | XXX |
| 22- ≤24 | XXX |
| Sex | |
| Male | XXX (XX.X) |
| Female | XXX (XX.X) |
| Residential area | 144 AV 15 |
| Urban/suburban | XXX (XX.X) |
| Rural | XXX (XX.X) |
| Missing | XXX (XX.X) |
| Residential status | |
| Permanent residents | XXX (XX.X) |
| Temporary residents | XXX (XX.X) |
| Missing | XXX (XX.X) |
| Birthweight [n (%)] | |
| Normal | XXX (XX.X) |
| Low birth weight | XXX (XX.X) |
| high birth weight | XXX (XX.X) |
| Missing | XXX (XX.X) |
| Gestational Age | |
| Full term | XXX (XX.X) |
| Pre-mature | XXX (XX.X) |
| Post-mature | XXX (XX.X) |

| Yes | XXX (XX.X) |
|-----------------------------------------------|------------|
| No | XXX (XX.X) |
| History of other seizures | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| History of febrile seizure | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| History of urticaria | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| History of angioedema | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| History of apnea | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| Fever at the date prior to 13vPnC vaccination | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |

<sup>\*</sup>Definition of baseline: Period between the 1st date of healthcare record (combining EHR and vaccination data) during the study period and 1st date of available 13vPnC dose (index date) recorded

| | Overall<br>n (%) |
|------------------------------------------|------------------|
| Number of participants | XXX |
| Age at entering the study [month] | |
| Mean (SD) | XXX (XX.X) |
| Median | XXX |
| Minimum | XXX |
| Maximum | XXX |
| Age groups at entering the study (month) | |
| 0- ≤2 | XXX |
| 2- ≤4 | XXX |
| 4- ≤6 | XXX |
| 6- ≤8 | XXX |
| 8- ≤10 | XXX |
| 10-≤12 | XXX |
| 12- ≤14 | XXX |
| 14- ≤16 | XXX |
| 16-≤18 | XXX |
| 18- ≤20 | XXX |
| 20- ≤22 | XXX |
| 22- ≤24 | XXX |
| Sex [n (%)] | |
| Male | XXX (XX.X) |
| Female | XXX (XX.X) |
| Residential area | |
| Urban/suburban | XXX (XX.X) |
| Rural | XXX (XX.X) |
| Missing | XXX (XX.X) |
| Residential status | |
| Permanent residents | XXX (XX.X) |
| Temporary residents | XXX (XX.X) |
| Missing | XXX (XX.X) |
| Birthweight | |
| Normal | XXX (XX.X) |
| Low birth weight | XXX (XX.X) |
| Gestational Age | |
| Full term | XXX (XX.X) |
| Pre-mature | XXX (XX.X) |

| Yes | XXX (XX.X) |
|-----------------------------------------------|------------|
| | XXX (XX.X) |
| No | max (max) |
| Sickle cell disease | VVV (VV V) |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| History of other seizures | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| History of febrile seizure | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| History of urticaria | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| History of angioedema | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| History of apnea | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| Fever at the date prior to 13vPnC vaccination | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |
| Smoking in the family | |
| Yes | XXX (XX.X) |
| No | XXX (XX.X) |

<sup>\*</sup>Definition of baseline: Period between the 1st date of healthcare record (combining EHR and vaccination data) during the Prospective cohort study period and 1st 13vPnC dose date

| | <b>Dose 1</b> n (%) | <b>Dose 2</b><br>n (%) | <b>Dose 3</b> n (%) | <b>Dose 4</b> n (%) |
|---|---|---|---|---|
| otal number of Participants | XXX | XXX | XXX | XXX |
| ge at each dose [month] | | | | |
| 0- ≤1 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 1- ≤2 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 2- ≤3 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 3- ≤4 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 4- ≤5 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 5- ≤6 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 6- ≤7 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 7- ≤8 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 8- ≤9 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 9- ≤10 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 10- ≤11 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 11-≤12 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 12-≤13 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 13- ≤14 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 14- ≤15 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 15- ≤16 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 16- ≤17 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 17-≤18 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 18- ≤19 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 19- ≤20 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 20- ≤21 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 21- ≤22 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 22- ≤23 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 23- ≤24 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
|---|---|---|---|---|
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Febrile seizures | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Urticaria and angioedema | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Apnea | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Fever | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Season of each dose | | | | |
| Winter (12/1-2/28) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Spring (3/1-5/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Summer (6/1-8/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Fall (9/1/-11/30) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year of administration | | | | |
| Year 1 (5/1/2017-4/30/2018) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year 2 (5/1/2018-4/30/2019) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year 3 (5/1/2019-7/24/2020) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Co-administration of other vaccines on the same date | | | | |
| Vaccine 1 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Vaccine 2 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |


| Vaccine 3 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
|---|---|---|---|---|
| Vaccine 4 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Vaccine 5 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Vaccine 6 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Table 2.2 Administration of 13vPnC by Dose - Prospect | ive Cohort Study | | | |
| | Dose 1 | Dose 2 | Dose 3 | Dose 4 |
| | n (%) | n (%) | n (%) | n (%) |
| Fotal number of Participants | XXX | XXX | XXX | XXX |
| Age at each dose [month] | | | | |
| 0- ≤1 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 1-≤2 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 2-≤3 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 3- ≤4 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 4- ≤5 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 5- ≤6 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 6- ≤7 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 7- ≤8 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 8- ≤9 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 9- ≤10 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 10-≤11 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 11-≤12 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 12- ≤13 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 13- ≤14 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 14-≤15 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 15-≤16 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 16- ≤17 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 17-≤18 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 18-≤19 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 19- ≤20 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 20- ≤21 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |

| 21-≤22 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
|---|---|---|---|---|
| 22-≤23 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 23-≤24 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Cety outcomes of interest and Hospitalization within | n 7 days of each dose | | | |
| All seizures | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Febrile Seizures | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Urticaria and angioedema | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Apnea | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Fever (≥38°C) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalized | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Highest temperature for each day fever is reported | | | | |
| Day 0 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Day 1 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Day 2 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Day 3 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |

| Day 4 | | | | |
|---|---|---|---|---|
| Day 5 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Day 6 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Day 7 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Fever* | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Season of each dose | | | | |
| Winter (12/1-2/28) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Spring (3/1-5/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Summer (6/1-8/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Fall (9/1/-11/30) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year of administration of 13vPnC | | | | |
| Year 1 (7/1/2018-6/30/2019) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year 2 (7/1/2019-7/24/2020) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Co-administration of other vaccines on the same date | | | | |
| Vaccine 1 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Vaccine 2 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Vaccine 3 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Vaccine 4 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Vaccine 5 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Vaccine 6 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Use of antipyretics post-vaccination within 7 days of each dose | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Use of concomitant drugs within 7 days of each dose | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |

<sup>\*</sup>Including those who had fever and reported temperature was greater than or equal to 38°C and those who had fever but not reported temperature "Participants didn't respond to the follow-up questionnaire on the seventh day after vaccination

Table 3.1 Distribution of Safety Outcomes of Interest\* - Main Study

| | | All Dose | | | | Dose 1 | | | Dose 2 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | All Seizures<br>n (%) | Urticaria and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>n (%) | All Seizures<br>n (%) | Urticaria and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>n (%) | All Seizures<br>n (%) | Urticaria and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>n (%) |
| Total number of Participants | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Age at 1st diagnosis [month] | | | | | | | | | | | | |
| Mean (SD) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Median | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Minimum | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Maximum | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Age at 1st diagnosis [month] | | | | | | | | | | | | |
| 0- ≤2 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2- ≤4 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4- ≤6 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6- ≤8 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8- ≤10 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10- ≤12 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12- ≤14 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 14- ≤16 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16- ≤18 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 18- ≤20 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20- ≤22 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 22- ≤24 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Sex | | | | | | | | | | | | |
| Male | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Female | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Residential area at study entry | | | | | | | | | | | | |
| Urban/suburban | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |

| Rural | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Residential status at study entry | | | | | | | | | | | | |
| Permanent residents | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Temporary residents | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalization within 7 days of each dose# | | | | | | | | | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Season of 1st diagnosis of each dose | | | | | | | | | | | | |
| Winter (12/1-2/28) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Spring (3/1-5/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Summer (6/1-8/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Fall (9/1/-11/30) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year of administration of 13vPnC associated with the | 1st diagnosis of each dose | | | | | | | | | | | |
| Year 1 (5/1/2017-4/30/2018) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year 2 (5/1/2018-4/30/2019) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year 3 (5/1/2019-7/24/2020) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |

<sup>\*</sup>Each outcome is within 7 days on or after each dose

<sup>\*</sup>A patient could be hospitalized after each dose, but the patient count would be 1

Table 3.1 Distribution of Safety Outcomes of Interest - Main Study

| | | Dose 3 | 3 | | T | Do | se 4 | |
|---|---|---|---|---|---|---|---|---|
| | All Seizures<br>n (%) | Urticaria and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>n (%) | All Seizures<br>n (%) | Urticaria and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>n (%) |
| Total number of Participants | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Age at 1st diagnosis [month] | | | | | | | | |
| Mean (SD) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Median | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Minimum | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Maximum | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Age at 1st diagnosis [month] | | | | | | | | |
| 0-≤2 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2-≤4 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4- ≤6 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6- ≤8 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8-≤10 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10-≤12 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12- ≤14 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 14- ≤16 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16- ≤18 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 18- ≤20 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20- ≤22 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 22- ≤24 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| ex | | | | | | | | |
| Male | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X |
| Female | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X |
| Residential area at study entry | | | | | | | | |
| Urban/suburban | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X |

## Statistical Analysis Plan

| Rural | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
|---|---|---|---|---|---|---|---|---|
| Residential status at study entry | | | | | | | | |
| Permanent residents | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Temporary residents | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Hospitalization within 7 days of each dose# | | | | | | | | |
| Yes | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| No | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Season of 1st diagnosis of each dose | | | | | | | | |
| Winter (12/1-2/28) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Spring (3/1-5/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Summer (6/1-8/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Fall (9/1/-11/30) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year of administration of 13vPnC associated with the 1st dia | gnosis of each dose | | | | | | | |
| Year 1 (5/1/2017-4/30/2018) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year 2 (5/1/2018-4/30/2019) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Year 3 (5/1/2019-7/24/2020) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |

<sup>\*</sup>Each outcome is within 7 days on or after each dose

<sup>#</sup>A patient could be hospitalized after each dose, but the patient count would be 1

Table 3.2 Distribution of Safety Outcomes of Interest\* - Prospective Cohort Study

| | | | All Dose | | | | | | Dose 1 | | | | | | Dose 2 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | All<br>seizures<br>n (%) | Febrile<br>seizures<br>n (%) | Urticaria<br>and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>(≥38°C)<br>n (%) | Highest temperature for each day fever is reported (≥39°C) n (%) | All<br>seizures<br>n (%) | Febrile<br>seizures<br>n (%) | Urticaria<br>and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>(≥38°C)<br>n (%) | Highest temperature for each day fever is reported (≥39°C) n (%) | | Febrile<br>seizures<br>n (%) | Urticaria<br>and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>(≥38°C)<br>n (%) | () |
| tal number of Participants | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | _ |
| ge at 1st diagnosis [month] | | | | | | | | | | | | | | | | | | _ |
| Mean (SD) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | ) XXX (XX.X) | XXX (XX.X) | ) XXX (XX.X) | A) |
| Median | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| Minimum | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| Maximum | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | _ |
| ge at 1st diagnosis [month] | | | | | | | | | | | | | | | | | | • |
| 0- ≤2 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 2- ≤4 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 4- ≤6 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 6- ≤8 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 8- ≤10 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 10-≤12 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 12-≤14 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 14- ≤16 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 16-≤18 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 18-≤20 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 20-≤22 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | |
| 22- ≤24 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | - |
| | | | | | | ļ | | | | | | ļ | | | | | | |
| Male | , , | XXX (XX.X) | , , | , , | | , , | ` ′ | , , | ` ' | , , | * * | , , | , , | XXX (XX.X) | , , , | , | , | |
| Female | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | ) XXX (XX.X) | XXX (XX.X) | XXX (XX. | У |

| Urb | pan/suburban | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Rura | ral | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Residential status at s | study entry | | | | | | | | | | | | | | | | | | |
| Perr | manent residents | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Ten | mporary residents | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Hospitalization within | n 7 days of each dose | | | | | | | | | | | | | | | | | | |
| Yes | S | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| No | | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Season of 1st diagnosi | is of each dose | | | | | | | | | | | | | | | | | | |
| Win | nter (12/1-2/28) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Spri | ing (3/1-5/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Surr | mmer (6/1-8/31) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Fall | 1 (9/1/-11/30) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Year of administratio with the 1st diagnosis | on of 13vPnC associated s of each dose | | | | | | | | | | | | | | | | | | |
| Yea | ar 1 (5/1/2017-4/30/2018) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Yea | ar 2 (5/1/2018-4/30/2019) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |
| Yea | ar 3 (5/1/2019-7/24/2020) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XX |

<sup>\*</sup>Each outcome is within 7 days on or after each dose

Table 3.2 Distribution of Safety Outcomes of Interest\* - Prospective Cohort Study

| | | | Dose 3 | | | | | | Dose 4 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | All seizures<br>n (%) | Febrile<br>seizures<br>n (%) | Urticaria<br>and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>(≥38°C)<br>n (%) | Highest<br>temperature<br>for each day<br>fever is<br>reported<br>(≥39°C)<br>n (%) | All<br>seizures<br>n (%) | Febrile<br>seizures<br>n (%) | Urticaria<br>and<br>angioedema<br>n (%) | Apnea<br>n (%) | Fever<br>(≥38°C)<br>n (%) | Highest<br>temperatur<br>for each da<br>fever is<br>reported<br>(≥39°C)<br>n (%) |
| Total number of<br>Participants | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Age at 1st diagnosis month] | | | | | | | | | | | | |
| Mean (SD) | XXX (XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X |
| Median | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Minimum | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Maximum | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Age at 1st diagnosis<br>month] | | | | | | | | | | | | |
| 0- ≤2 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2- ≤4 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4- ≤6 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6- ≤8 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8-≤10 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10-≤12 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12-≤14 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 14- ≤16 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16-≤18 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 18-≤20 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20-≤22 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 22-≤24 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| ex | | | | | | | | | | | | |
| Male | XXX (XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X |
| Female | XXX (XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | (XXX) | XXX<br>(XX.X) | XXX (XX.X |

| _ | | | | | | | _ | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Urban/suburban | XXX (XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) |
| Orban/suburban | | XXX | | XXX | XXX | | XXX | XXX | | XXX | XXX | |
| Rural | XXX (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) |
| Residential status at | | | | | | | | | | | | |
| study entry | | 3/3/3/ | | NAVA. | 3/3/3/ | | 3/3/3/ | 3/3/3/ | | 373737 | 373737 | |
| Permanent<br>residents | XXX (XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) |
| Temporary | | XXX | | XXX | XXX | | XXX | XXX | | XXX | XXX | |
| residents | XXX (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) |
| Hospitalization | | | | | | | | | | | - | |
| within 7 days of | | | | | | | | | | | | |
| each dose | | 373737 | | 77777 | 373737 | | 3/3/3/ | ***** | | 373737 | 373737 | |
| Yes | XXX (XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) |
| | | XXX | | XXX | XXX | | XXX | XXX | | XXX | XXX | |
| No | XXX (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) |
| Season of 1st | | , , | | , | , | | | , , | | ` ' | , | |
| diagnosis of each | | | | | | | | | | | | |
| dose | | 373737 | | 77777 | ***** | | 3/3/3/ | 373737 | | 373737 | 373737 | |
| Winter (12/1-<br>2/28) | XXX (XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) | XXX<br>(XX.X) | XXX<br>(XX.X) | XXX (XX.X) |
| Spring (3/1- | | XXX | | XXX | XXX | | XXX | XXX | | XXX | XXX | |
| 5/31) | XXX (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) |
| Summer (6/1- | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX | VVV (VV V) | XXX | XXX | XXX (XX.X) | XXX | XXX | VVV (VV V) |
| 8/31) | ΛΛΛ (ΛΛ.Λ) | (XX.X) | ΛΛΛ (ΛΛ.Λ) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda)$ | (XX.X) | (XX.X) | XXX (XX.X) |
| Fall (9/1/- | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX | XXX (XX.X) | XXX | XXX | XXX (XX.X) | XXX | XXX | XXX (XX.X) |
| 11/30) | | (XX.X) | | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | | (XX.X) | (XX.X) | · / |
| Year of administration of | | | | | | | | | | | | |
| 13vPnC associated | | | | | | | | | | | | |
| with the 1st | | | | | | | | | | | | |
| diagnosis of each | | | | | | | | | | | | |
| dose | | | | | | | | | | | | |
| Year 1 | 77777 (7777 X** | XXX | van an v | XXX | XXX | 17777 A777 T | XXX | XXX | 17171 (1717 T | XXX | XXX | 77777 (7777 7° |
| (5/1/2017-<br>4/30/2018) | XXX (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) |
| 4/30/2018)<br>Year 2 | | | | | | | | | | | | |
| (5/1/2018- | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX | XXX (XX.X) | XXX | XXX | XXX (XX.X) | XXX | XXX | XXX (XX.X) |
| 4/30/2019) | ( | (XX.X) | ( | (XX.X) | (XX.X) | () | (XX.X) | (XX.X) | () | (XX.X) | (XX.X) | ( |
| Year 3 | | XXX | | XXX | XXX | | XXX | XXX | | XXX | XXX | |
| (5/1/2019- | XXX (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) | (XX.X) | (XX.X) | XXX (XX.X) |
| 7/24/2020) | | (2121.21) | | (222.21) | (222.21) | | (222.22) | (222.21) | | (222.22) | (2121.21) | |

<sup>\*</sup>Each outcome is within 7 days on or after each dose.

| | | Dose 1 ( | 0-3 days) | | Dose 1 ( | 4-7 days) | | Dose 1 | (0-7 days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 ( | 0-3 days) | | Dose 2 ( | 4-7 days) | | Dose 2 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 ( | (0-3 days) | | Dose 3 ( | 4-7 days) | | Dose 3 | (0-7 days) |
| | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | s (0-3 days) | | All Doses | s (4-7 days) | | All Dose | es (0-7 days) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| angioedema | ΛΛΛ | 717171 | AA:A(AA:A - AA:A) | 717171 | 71271 | 721.71 (721.71 721.71) | | | , |

| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|

| | | | | Age 0- ≤2 r | nonths | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | Dose 1 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 days) | | | | Dose 2 (4-7 days) | | | lays) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Dose 3 (0-3 days) Dose 3 (4-7 days) Dose 3 (0-7 days)

| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0- | -3 days) | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |
| P | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events All seizures | XXX | XXX | NA A AN A NA NA | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 2- ≤4 1 | months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 c | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at risk (n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 c | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at risk (n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ |
| | | | . , , | | | | | | |
| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 o | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0- | -3 days) | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 4- ≤6 ı | months | | | | |
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 c | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of<br>events<br>(n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
|---|---|---|---|---|---|---|---|---|---|
| | Dose 4 (0-3 days) | | | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | lays) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | lays) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 days) | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| All seizures<br>Febrile seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0- | -3 days) | | All Doses (4- | 7 days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 6- ≤8 ı | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | days) | Dose 1 (4-7 days) | | | | Dose 1 (0-7 c | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 c | lays) |

| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
|---|---|---|---|---|---|---|---|---|---|
| Events | | | | | | | | | <u> </u> |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 c | lays) |
| _ | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events | XXX | VVV | | XXX | XXX | VV V (VV V VV V) | XXX | XXX | VV V (VV V VV V) |
| All seizures | | XXX | XX.X (XX.X - XX.X) | | | XX.X (XX.X - XX.X) | | | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 c | lays) |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4- | 7 days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 8- ≤10 | months | | | | |
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | Dose 1 (0-7 days) | | |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 c | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |


| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 c | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | days) | Dose 4 (4-7 days) | | | | Dose 4 (0-7 days) | |
| | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events | | | | | | | | | <u> </u> |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Urticaria and

angioedema

Apnea

Fever

XXX

XXX

XXX

XXX

XXX

XXX

| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

## Age 10-≤12 months Dose 1 (0-3 days) Dose 1 (4-7 days) Dose 1 (0-7 days) Number of Person days Number of Person days Incidence Rate per Number of Person days at Incidence Rate per **Incidence Rate per 1000** 1000 person days (95% at risk at risk 1000 person days (95% risk events events events person days (95% CI) (n) (n) (n) (n) CI) (n) (n) CI) **Events** All seizures XXX XXXXXXXXXXX.X (XX.X - XX.X) XXX XXXXX.X (XX.X - XX.X) XX.X (XX.X - XX.X) Febrile seizures XXX XXXXXX XXX XX.X (XX.X - XX.X) XXX XXXXX.X (XX.X - XX.X) XX.X (XX.X - XX.X) Urticaria and XXXXXXXXXXXXXX.X(XX.X - XX.X)XXXXXXXX.X (XX.X - XX.X) angioedema XX.X (XX.X - XX.X) XXXApnea XXXXXXXXXXX.X (XX.X - XX.X) XXXXXX XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XXXXXXXXXXXX XX.X(XX.X - XX.X)XXX XXXXX.X (XX.X - XX.X) Fever XX.X(XX.X - XX.X)Dose 2 (0-3 days) Dose 2 (4-7 days) Dose 2 (0-7 days) Number of Person days Incidence Rate per Number of Person days at Incidence Rate per Person days Number of Incidence Rate per 1000 events at risk at risk 1000 person days (95% risk 1000 person days (95% events events person days (95% CI) (n) (n) (n) (n) CI) (n) (n) CI) **Events** All seizures XX.X (XX.X - XX.X) XXXXX.X (XX.X - XX.X) XXX XXXXXXXXX XXX XX.X (XX.X - XX.X) Febrile seizures XXXXXXXXXXXXXXX XX.X (XX.X - XX.X) XXXXX.X(XX.X - XX.X)XX.X(XX.X - XX.X)

XX.X(XX.X - XX.X)

XX.X(XX.X - XX.X)

XX.X(XX.X - XX.X)

XXX

XXX

XXX

XXX

XXX

XXX

XX.X (XX.X - XX.X)

XX.X (XX.X - XX.X)

XX.X (XX.X - XX.X)

XXX

XXX

XXX

XXX

XXX

XXX

XX.X (XX.X - XX.X)

XX.X (XX.X - XX.X)

XX.X (XX.X - XX.X)

| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | lays) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0- | -3 days) | | All Doses (4- | -7 days) | | All Doses (0-7 | days) |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 12- ≤14 | months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 d | lays) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at risk (n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 c | lays) |
| | | | | Age 14- ≤16 | months | | | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| | All Doses (0-3 days) | | | | All Doses (4- | -7 days) | | All Doses (0-7 | days) |
| | | | | | | , | | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| angioedema Apnea | XXX<br>XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) |
| Febrile seizures Urticaria and | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of<br>events<br>(n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 c | lays) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of<br>events<br>(n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
|---|---|---|---|---|---|---|---|---|---|
| | | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | lays) | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | lays) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 | days) | Dose 2 (0-7 days) | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| All seizures<br>Febrile seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0- | -3 days) | | All Doses (4- | 7 days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | Dose 1 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 c | lays) |

| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | lays) |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events All seizures | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ |
| | λλλ | λλλ | XX.X (XX.X - XX.X) | λλλ | АЛА | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ | λλλ | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | lays) |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events | | | | | | | | | · |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4- | 7 days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 18- ≤20 | months | | | | |
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 d | lays) |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 d | lays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |


| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 | days) | Dose 3 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | days) | Dose 4 (4-7 days) | | | | Dose 4 (0-7 o | lays) |
| | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events | | | | | | | | | , |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0- | -3 days) | | All Doses (4- | 7 days) | All Doses (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

## Age 20- ≤22 months Dose 1 (0-3 days) Dose 1 (4-7 days) Dose 1 (0-7 days) Number of Person days Number of Person days Incidence Rate per Number of Person days at Incidence Rate per **Incidence Rate per 1000** 1000 person days (95% 1000 person days (95% at risk at risk risk events events events person days (95% CI) (n) (n) (n) (n) CI) (n) (n) CI) **Events** XXXXX.X (XX.X - XX.X) XX.X (XX.X - XX.X) All seizures XXX XXXXXX XXXXXXXX.X (XX.X - XX.X) XXX XXX XX.X (XX.X - XX.X) Febrile seizures XXXXXX XXX XXXXX.X (XX.X - XX.X) XX.X (XX.X - XX.X) Urticaria and XXX XX.X (XX.X - XX.X) XXXXXXXXX XXXXXXXX.X (XX.X - XX.X) angioedema XX.X (XX.X - XX.X) XXXXXX XXX XXXApnea XXXXXX XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) Fever XXX XXXXXXXXX XX.X (XX.X - XX.X) XXXXXXXX.X (XX.X - XX.X) XX.X (XX.X - XX.X)

| | | Dose 2 (0-3 | days) | <b>Dose 2 (4-7 days)</b> | | | Dose 2 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Dose 3 (0-3 days) Dose 3 (4-7 days) Dose 3 (0-7 days)

| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 days) | | | Dose 4 (0-7 days) | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | All Doses (4-7 days) | | | All Doses (0-7 days) | | |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| Events All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 22- ≤24 | months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 days) | | | Dose 1 (0-7 days) | |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 | days) | Dose 3 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 4 (0-3 days) | | | Dose 4 (4-7 days) | | | Dose 4 (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0- | -3 days) | | All Doses (4-7 days) | | | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|--|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days (95%<br>CI) | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| | | | | Male | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 | (0-3 days) | | Dose 1 (4-7 | days) | | Dose 1 | (0-7 days) |
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | | Dose 2 | (0-3 days) | | Dose 2 (4-7 | days) | | Dose 2 | (0-7 days) |
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |

| Events | Number of events (n) | Person<br>months at risk<br>(n) | Incidence Rate per 1,000 person<br>months (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | a XXX XXX XXX XX.X (XX.X - XX.X) | | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 4 (0-3 days) | | | | Dose 4 (4-7 | ' days) | Dose 4 (0-7 days) | | |
| Events | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | es (0-3 days) | | All Doses (4- | -7 days) | | All Dose | s (0-7 days) |
| Events | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX XXX XX.X (XX.X - XX.X) | | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | | | | Female | | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 days) | |
| P | Number of events (n) | Person days at risk (n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| Events All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | | Dose 2 | (0-3 days) | | days) | Dose 2 (0-7 days) | | | |
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |

| | | Dose 3 | (0-3 days) | | Dose 3 (4-7 | days) | Dose 3 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person<br>months at risk<br>(n) | Incidence Rate per 1,000 person<br>months (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number of events (n) Person days at risk (n) | | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 (4-7 | days) | Dose 4 (0-7 days) | | |
| Г | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | es (0-3 days) | | All Doses (4- | 7 days) | | All Dose | s (0-7 days) |
| Events | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| NIS Protocol | <b1851193></b1851193> |
|--------------|-----------------------|

## Statistical Analysis Plan

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | Permanent | residents | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 da | ays) | | Dose 1 (4-7 da | Dose 1 (0-7 days) | | | |
| Events | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | | Dose 2 (0-3 da | ays) | | Dose 2 (4-7 da | nys) | | Dose 2 | (0-7 days) |
| Events | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX. |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX. |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |

| Events | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 da | ays) | | Dose 4 (4-7 da | | Dose 4 | (0-7 days) | |
| Events | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0-3 | days) | | All Doses (4-7 d | lays) | | All Dose | s (0-7 days) |
| Events | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
|---|---|---|---|---|---|---|---|---|
| XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | | Temporary | residents | | | | | |
| | Dose 1 (0-3 da | ays) | | Dose 1 (4-7 da | nys) | | Dose 1 | (0-7 days) |
| Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | Dose 2 (0-3 da | ays) | | | | (0-7 days) | | |
| Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| ΛΛΛ | AAA | | | | | | | |
| XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | Number of events (n) XXX XXX XXX XXX XXX XXX XXX | Number of events (n) Number of events (n) XXX XXX XXX XXX XXX XXX XXX XX | Number of events (n) | XXX | Number of events (n) | Number of events (n) Dose 1 (0-3 days) Dose 2 (0-3 days) D | Number of events (n) | XXX |

| | | Dose 3 (0-3 da | ays) | | Dose 3 (4-7 da | ays) | Dose 3 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 days) | | | Dose 4 (4-7 days) | | | Dose 4 (0-7 days) | |
| Events | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk (n) | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0-3 | days) | | All Doses (4-7 o | days) | | All Dose | es (0-7 days) |
| Events | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person days at risk | Incidence Rate per<br>1,000 person days<br>(95%CI) | Number<br>of<br>events<br>(n) | Person<br>days<br>at risk<br>(n) | Incidence Rate per<br>1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Table 4.1.5 Incidence Rates (Per 1000 person days) of Safety Outcomes of Interest - Main Study (by Co-administration of other vaccines on the same date)

| | | | Co-administrat | ion of other vacc | ines on the same o | date (Yes)* | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 c | days) | Dose 1 (0-7 days) | | |
| T. | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | , | | | ` ' | | | ` ′ |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 d | lays) | Dose 2 (0-7 days) | | |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| Events | ****** | ****** | ****************************** | ****** | ****** | ****** | ****** | 77777 | ***************** |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 d | lays) | Dose 3 (0-7 days) | | |
| Evente | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 d | lays) | Dose 4 (0-7 days) | | |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0- | -3 days) | | All Doses (4-7 | days) | | All Doses (0-7 | days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| I III SCIZUICS | | | | | | | | | |

| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 d | lays) | Dose 1 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 d | lays) | | Dose 2 (0-7 d | ays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |

| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 d | lays) | | Dose 4 (0-7 d | ays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0- | -3 days) | | All Doses (4-7 | ' days) | | All Doses (0-7 | days) |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| Events | ***** | ****** | | ****** | ****** | *************************************** | ****** | ****** | ************* |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

<sup>\*</sup>Any dose of 13vPnC has been vaccinated on the same day as the other vaccines.

| | | | | | Winter | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 | (4-7 days) | | Dose 2 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of<br>events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | 4 (4-7 days) | | Dose 4 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dos | es (0-3 days) | | All Dos | es (4-7 days) | | All Dose | s (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| NIS Protocol | <b1851193></b1851193> |
|--------------|-----------------------|

## Statistical Analysis Plan

| | Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| ] | Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | Dose 1 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | 2 (0-3 days) | | Dose 2 | 2 (4-7 days) | | Dose 2 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | 6 (0-3 days) | | Dose 3 | 8 (4-7 days) | | Dose 3 | (0-7 days) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | 4 (0-3 days) | | Dose 4 | 4 (4-7 days) | | Dose 4 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of<br>events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dos | es (0-3 days) | | All Dos | es (4-7 days) | | All Dose | s (0-7 days) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| angioedema | | | ` ′ | | | ` / | | | |

| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Summer | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | 2 (0-3 days) | | Dose 2 | 2 (4-7 days) | | | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | (0-3 days) | | Dose 3 | 6 (4-7 days) | | Dose 3 | (0-7 days) |

| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | 4 (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 | (0-7 days) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | All Dos | es (4-7 days) | | All Dose | s (0-7 days) | |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| All Seizures Febrile seizures | xxx<br>xxx | xxx<br>xxx | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | xxx<br>xxx | xxx<br>xxx | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,00<br>person days (95%CI) |
| | | Dose 2 | 2 (0-3 days) | | Dose 2 | (4-7 days) | | Dose 2 | (0-7 days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,00<br>person days (95%CI) |
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | Dose 1 (0-7 days) | | |
| | | | | | Fall | | | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| ngioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 3 | 3 (0-3 days) | | Dose 3 | 3 (4-7 days) | | Dose 3 | (0-7 days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | 4 (0-3 days) | | Dose 4 | l (4-7 days) | Dose 4 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dos | es (0-3 days) | | All Dos | es (4-7 days) | | All Dose | s (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 | (0-3 days) | | Dose 1 (4- | 7 days) | | Dose 1 ( | 0-7 days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 (4- | 7 days) | Dose 2 (0-7 days) | | |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | (0-3 days) | | Dose 3 (4- | 7 days) | | Dose 3 ( | 0-7 days) |
| | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 (4- | 7 days) | | Dose 4 ( | 0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses | s (0-3 days) | | All Doses (4 | 1-7 days) | | All Doses | (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| angioedema | | | | | | | | | |


| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|

| | | | | Age 0- ≤ | 2 months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | ys) | | Dose 2 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Dose 3 (0-3 days) Dose 3 (4-7 days) Dose 3 (0-7 days)

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Events | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0 | )-3 days) | | All Doses (4-7 d | ays) | | All Doses (0- | 7 days) |
| F | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | WWW WWW WWW | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 2- ≤ | 4 months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | | Dose 1 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | ys) | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 4- <u></u> | ≤6 months | | | | |
| | | Dose 1 (0- | 3 days) | | Dose 1 (4-7 da | ys) | | Dose 1 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |


| | Number of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 4 (0- | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| | | Dose 3 (0- | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| | | Dose 2 (0-2 | 3 days) | | Dose 2 (4-7 da | ys) | | Dose 2 (0-7 | days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| All seizures<br>Febrile seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | | All Doses (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 (0-3 | 3 days) | 9 - | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| F.,4- | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses<br>(n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 da | vs) | | Dose 2 (0-7 | days) |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | Number of events (n) Number of doses (n) Number of total Incidence Rate per 1,000 doses (95% CI | | |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | events | doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | VVV | | VVV | XXX | VV V (VV V VV V) | | VVV | VVV (VV V VVV) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 8- ≤ | 10 months | | | | |
| | Dose 1 (0-3 days) | | | | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
| T | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses<br>(n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | VV V AVV V VV V | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | ys) | | Dose 2 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |


| A | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | ` ′ | XXX | XXX | ` ′ |
| Fever | λλλ | AAA | XX.X (XX.X - XX.X) | AAA | XXX | XX.X (XX.X - XX.X) | λλλ | AAA | XX.X (XX.X - XX.X |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da) | ys) | Dose 3 (0-7 days) | | |
| Events | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0 | 3 days) | | Dose 4 (4-7 da) | ys) | | Dose 4 (0-7 days) | |
| T | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0 | )-3 days) | | All Doses (4-7 d | ays) | | All Doses (0- | 7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| A 00 1 | 0 /12 | months |
|--------|----------|--------|
| Age II | U- < I Z | months |

| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | | Dose 1 (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |

| | | Dose 2 (0-3 days) | | | Dose 2 (4-7 da | ys) | | Dose 2 (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Dose 3 (0-3 days) Dose 3 (4-7 days) Dose 3 (0-7 days)
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0 | )-3 days) | | All Doses (4-7 d | ays) | | All Doses (0-7 | 7 days) |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | VVV | VVV | | VVV | VVV | VV V (VV V VV V) | VVV | VVV | VV V (VV V VV V) |
| All seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | λλλ | λλλ | XX.X (XX.X - XX.X) | λλλ | λλλ | XX.X (XX.X - XX.X) | λλλ | λλλ | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 12- ≤ | 14 months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da) | ys) | | Dose 1 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0 | 3 days) | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0- | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | | Dose 1 (0-7 | days) |
| | | | | Age 14- ≤ | 16 months | | | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | | All Doses (0- | 7 days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| angioedema Apnea | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) |
| Febrile seizures Urticaria and | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of<br>events<br>(n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of<br>events<br>(n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | Number of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| | Dose 4 (0-3 days) | | | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| | | Dose 3 (0- | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| | | Dose 2 (0-2 | 3 days) | | Dose 2 (4-7 da | ys) | | Dose 2 (0-7 | days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| All seizures Febrile seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | vs) | | Dose 2 (0-7 | davs) |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | VVV | | VVV | VVV | VV V (VV V VV V) | | VVV | VVV (VV V VVV) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses<br>(n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 18- ≤ | 20 months | | | | |
| | Dose 1 (0-3 days) | | | | Dose 1 (4-7 da) | ys) | Dose 1 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0 | 3 days) | | Dose 2 (4-7 da) | ys) | | Dose 2 (0-7 | days) |
| Events | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |


| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0- | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0- | 3 days) | Dose 4 (4-7 days) | | | Dose 4 (0-7 days) | | |
| | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | | | | 3/3/3/ | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | | All Doses (4-7 d | lays) | | All Doses (0- | 7 days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

## Age 20- ≤22 months

| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | Dose 2 (0-3 days) | | | | Dose 2 (4-7 da | ys) | Dose 2 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0 | )-3 days) | | All Doses (4-7 d | ays) | | All Doses (0-7 | 7 days) |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | VVV | VVV | | VVV | VVV | VV V (VV V VV V) | VVV | VVV | VV V (VV V VV V) |
| All seizures Febrile seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
| | ΛΛΛ | ΛΛΛ | XX.X (XX.X - XX.X) | ΛΛΛ | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ | ΛΛΛ | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 22-≤ | 24 months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | | Dose 1 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | ys) | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | Dose 4 (0-3 days) | | | | Dose 4 (4-7 da | ys) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | All Doses (0-3 days) | | | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | N. | lale | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 | (0-3 days) | | Dose 1 (4- | 7 days) | Dose 1 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 (4- | 7 days) | | Dose 2 ( | 0-7 days) |
| Events | (n) (n) (95%CI) | | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 (4- | 7 days) | | Dose 4 ( | 0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | s (0-3 days) | | All Doses ( | 1-7 days) | | All Doses | (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Female | | | | | | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 (4- | -7 days) | | Dose 1 ( | 0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,00<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 (4- | -7 days) | | Dose 2 ( | 0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,00<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 3 | (0-3 days) | | Dose 3 (4- | -7 days) | Dose 3 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | Dose 4 (4-7 days) | | | Dose 4 (0-7 days) | | |
| Events | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | s (0-3 days) | | All Doses ( | 4-7 days) | | All Doses | (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |

| | | | | Peri | manent residents | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | De | ose 1 (0-3 days) | | Dose 1 (4-7 days) | | | Dose 1 ( | (0-7 days) |
| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses<br>(n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | D | ose 2 (0-3 days) | | Dose 2 (4-7 days) | | | Dose 2 ( | (0-7 days) |
| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses<br>(n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | D | ose 4 (0-3 days) | | Dose 4 (4-7 days) | | | Dose 4 ( | 0-7 days) |
| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | All Doses (4-7 days) | | | All Doses | (0-7 days) | |
| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Temporary resident | ts | | | | | | | | |
| | | D | ose 1 (0-3 days) | | Dose 1 (4-7 days) | | | Dose 1 ( | (0-7 days) |
| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | D | ose 2 (0-3 days) | | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | |
| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | D | ose 3 (0-3 days) | | Dose 3 (4-7 days) | | Dose 3 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | D | ose 4 (0-3 days) | Dose 4 (4-7 days) | | | | Dose 4 | (0-7 days) |
| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | All Doses (4-7 days) | | | All Doses | s (0-7 days) | |
| Events | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number<br>of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number<br>of<br>events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Table 4.2.5 Incidence Rates | (Per 1000 Doses) of Safet | v Outcomes of Interest | - Main Study (by | Co-administration of other | r vaccines on the same date) |
|---|---|---|---|---|---|

| | | Dose 1 ( | 0-3 days) | | | Dose 1 (4-7 days) | | Dose 1 (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| E | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 2 (0-3 days) | | | | | Dose 2 (4-7 days) | Dose 2 (0-7 days) | | |
| | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |

| Events | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 3 ( | (0-3 days) | | | Dose 3 (4-7 days) | | Dose 3 (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 ( | (0-3 days) | | | Dose 4 (4-7 days) | Dose 4 (0-7 days) | | |
| Events | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses | s (0-3 days) | | | All Doses (4-7 days) | | All Doses (0-7 days | ) |
| Events | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Co-admin | stration of other vaccines on the same date (No) | | | |
| | | Dose 1 ( | 0-3 days) | | | Dose 1 (4-7 days) | Dose 1 (0-7 days) | | |
| Events | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 2 (0-3 days) | | | | | Dose 2 (4-7 days) | | Dose 2 (0-7 days) | |
| Fuonts | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 3 (0-3 days) | | | | | Dose 3 (4-7 days) | | Dose 3 (0-7 days) | |
| Events | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |


| | | Dose 4 | (0-3 days) | | | Dose 4 (4-7 days) | | Dose 4 (0-7 days | 3) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 4 ( | (0-3 days) | | | Dose 4 (4-7 days) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses | s (0-3 days) | | | All Doses (4-7 days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per<br>1,000 doses (95%<br>CI) | Number<br>of events<br>(n) | Number<br>of doses<br>(n) | Incidence Rate per 1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

<sup>\*</sup>Any dose of 13vPnC has been vaccinated on the same day as the other vaccines.

| | | | | | Winter | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 | (0-3 days) | Dose 1 (4-7 days) | | | Dose 1 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 2 (0-3 days) | | | | Dose 2 | (4-7 days) | | Dose 2 (0 | 9-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | (4-7 days) | Dose 4 (0-7 days) | | |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | s (0-3 days) | | All Dose | s (4-7 days) | | All Doses | (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | | Spring | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 (0 | -7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 | (4-7 days) | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | | | | | |


| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 3 | (0-3 days) | | Dose 3 | (4-7 days) | Dose 3 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 (0 | -7 days) |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | | All Doses (4-7 days) | | | All Doses (0-7 days) | |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | | Summer | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 (4-7 days) | | | Dose 1 (0 | -7 days) |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All Seizules | AAA | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ | ΛΛΛ | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ | ΛΛΛ | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 2 (0-3 days) | | | | Dose 2 | (4-7 days) | | Dose 2 (0 | -7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |

| | <u></u> | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | (0-3 days) | | Dose 3 | (4-7 days) | | Dose 3 (0 | )-7 days) |
| | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | )-7 days) | | | |
| Events | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | s (0-3 days) | | All Dose | es (4-7 days) | All Doses (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | | Fall | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 (4-7 days) | | | Dose 1 (0-7 days) | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | | | | Dose 2 (0-7 days) | | |

| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 3 (0-3 days) | | | | Dose 3 | (4-7 days) | Dose 3 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 4 (0-3 days) | | | | Dose 4 | (4-7 days) | | Dose 4 (0 | -7 days) |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | es (0-3 days) | | All Dose | s (4-7 days) | | All Doses | (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 | (0-7 days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 | 2 (4-7 days) | | Dose 2 (0-7 days) | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | (0-3 days) | | Dose 3 | 8 (4-7 days) | Dose 3 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
|---|---|---|---|---|---|---|---|---|---|--|
| | | Dose 4 | (0-3 days) | | Dose 4 | 4 (4-7 days) | | Dose 4 | (0-7 days) | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| | | All Dos | es (0-3 days) | | All Dos | es (4-7 days) | All Doses (0-7 days) | | | |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | |
| | | | | Age 0- ≤2 m | onths | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 d | lays) | | Dose 1 (4-7 | days) | Dose 1 (0-7 days) | | |
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 c | lays) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 d | ays) |
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | ****** | ****** | | ****** | ****** | *************************************** | 77777 | ****** | *************************************** |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 d | lays) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | ays) |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | NAME AND A STATE OF THE STATE O | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| 1111 BUIZUIUS | AAA | AAA | XX.X (XX.X - XX.X) | AAA | $\Lambda \Lambda \Lambda$ | AA.A(AA.A - AA.A) | MM | AAA | AA.A (AA.A - AA.A) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |

| pnea | XX.X - XX.X) $XXX$ $XXX$ $XX.X$ $(XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX$ | X.X - XX.X) |
|---|---|---|
| ever | XX.X - XX.X) XXX XXX XX.X (XX | X.X - XX.X) |
| | XX.X - XX.X) XXX XXX | ` |

| | | Dose 4 (0-3 c | lays) | | Dose 4 (4-7 | days) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0-3 | days) | All Doses (4-7 days) | | | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Age 2- ≤4 months

Dose 1 (0-3 days) Dose 1 (0-7 days)

| | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| Events | VVV | VVV | | VVV | VVV | VV V (VV V VV V) | VVV | VVV | VV V (VV V VV V) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 c | days) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 d | ays) |
| Forest | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 c | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | ays) |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 4 (0-3 d | lays) | | Dose 4 (4-7 | days) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0-3 | days) | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |
| | Number of events (n) | Person days at risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | | | | | (-) | | | | |
| All seizures | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 4- ≤6 m | onths | | | | |
| | | Dose 1 (0-3 o | lays) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 d | ays) |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 c | days) | | Dose 2 (4-7 | days) | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 3 (0-3 days) | | | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | ays) |
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | ***** | ***** | | ***** | | | ***** | ****** | ****************** |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 o | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | ays) |
| Б | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | NN N (NN N NN N | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and angioedema | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| - | | | XX.X (XX.X - XX.X) | | | | | | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0-3 | 3 days) | | All Doses (4-7 days) | | | All Doses (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 (0-3 o | lays) | | Dose 1 (4-7 days) | | | Dose 1 (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 o | lays) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 d | ays) |

| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| Events | | | | | (11) | | | | |
| All seizures | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 c | lays) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | lays) |
| P. A | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 o | lays) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | lays) |
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0-3 | days) | | All Doses (4- | 7 days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | WWW WWW WWW | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| reoffic scizures | ΛΛΛ | ΛΛΛ | XX.X (XX.X - XX.X) | λλλ | λλλ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ | АЛА | АЛА | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 8- ≤10 n | nonths | | | | |
| | Dose 1 (0-3 days) | | | | Dose 1 (4-7 | days) | Dose 1 (0-7 days) | | |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | AA.A (AA.A - AA.A) | | | , | | | |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 c | lays) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 da | ays) |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 ( | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | ays) |
| _ | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | VVV | VVV | | VVV | VVV | VV V (VV V VV V) | VVV | WWW | VV V (VV V VV V) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 o | lays) | Dose 4 (4-7 days) | | | | Dose 4 (0-7 d | ays) |
| Events | Number of events | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0-3 | days) | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | | | | | | | | | |
| | | | | | | | ***** | 373737 | 3737 37 (3737 37 3737 37) |
| All seizures Febrile seizures | XXX | XXX<br>XXX | XX.X (XX.X - XX.X) | XXX<br>XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and angioedema | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | XX.X(XX.X - XX.X) | | | | | | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 10- ≤12 r | nonths | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 ( | lays) | | Dose 1 (4-7 | days) | Dose 1 (0-7 days) | | |
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 c | days) | | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | |
| | Number of events | Person days at risk | Incidence Rate per 1000 person | Number of events | Person days at | Incidence Rate per 1000 person | Number of events | Person days at risk | Incidence Rate per 1000 person |

| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Dose 3 (0-3 days) Dose 3 (4-7 days)

| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 d | lays) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 da | ays) |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0-3 | days) | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 12- ≤14 r | months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 d | lays) | | Dose 1 (4-7 | days) | Dose 1 (0-7 days) | | |
| F4. | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 days) | | | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 c | lays) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | ays) |
| Frank | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 c | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | ays) |
| _ | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |
| т. | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 14- ≤16 r | nonths | | | | |
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 d | ays) |
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | MAN (MAN) | | | , | | | |

| Apnea<br>Fever | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | NN N (NN N NN N) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | ΛΛ.Λ (ΛΛ.Λ - ΛΛ.Λ) | | | ` ' | | | , |
| All seizures Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
| Events All seizures | XXX | XXX | | XXX | XXX | VV V (VV V VV V) | XXX | XXX | VV V (VV V VV V) |
| | Number of events (n) | Person days at risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| | | Dose 3 (0-3 c | lays) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | ays) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Person days at risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| | | Dose 2 (0-3 c | lays) | | Dose 2 (4-7 | days) | Dose 2 (0-7 days) | | |
| revei | AAA | AAA | XX.X (XX.X - XX.X) | AAA | AAA | ΛΛ.Λ (ΛΛ.Λ - ΛΛ.Λ) | AAA | AAA | ΛΛ.Λ (ΛΛ.Λ - ΛΛ.Λ) |
| Apnea<br>Fever | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| All seizures Febrile seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0-3 | 3 days) | | All Doses (4- | 7 days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | *************************************** | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | XX.X (XX.X - XX.X) | | | , | | | , |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| e e e e e e e e e e e e e e e e e e e | | | XX.X (XX.X - XX.X) | | | , | | | , |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | , | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Tever | AAA | ΛΛΛ | XX.X (XX.X - XX.X) | ΛΛΛ | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ | ΛΛΛ | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ |

| | | Dose 1 (0-3 d | lays) | Dose 1 (4-7 days) | | | Dose 1 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| Events | | | | | (n) | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 c | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | ays) |
| F. 4 | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 c | days) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | ays) |
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |

| | | All Doses (0-3 | days) | | All Doses (4- | 7 days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 18- ≤20 r | nonths | | | | |
| | | Dose 1 (0-3 o | lays) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 d | ays) |
| | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | VVV | | VVV | VVV | VV V (VV V VV V) | VVV | VVV | VV V (VV V VV VV |
| | | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 c | lays) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 d | ays) |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 c | lays) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | ays) |
| | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | NNN. | VVV | | VVV | XXX | WWW (WWW WWW) | VVV | VVV | VV V (VV V VV V) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 o | lays) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | ays) |
| Events | Number of events | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0-3 | days) | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |
| | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| T . | | | | | | | | | |
| Events | | | | | ** | | | | |
| All seizures Febrile seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |

| Urticaria and angioedema | XXX | XXX | | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | XX.X(XX.X - XX.X) | | | | | | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |

| | | | | Age 20- ≤22 ı | months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 | days) | Dose 1 (0-7 days) | | |
| | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 persor<br>days (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 d | ays) |

| | | D03C 2 (0-3 ( | iays) | | D03C 2 (4-7 | unjsj | Dose 2 (0-1 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Dose 3 (0-3 days) Dose 3 (4-7 days)

| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 d | lays) | | Dose 4 (4-7 | days) | | Dose 4 (0-7 d | ays) |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0-3 | days) | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |
| | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events | ****** | ***** | | ****** | ***** | | ***** | ***** | ******************* |
| All seizures | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 22- ≤24 r | nonths | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 d | lays) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 d | ays) |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | NA N WAY Y NA NA | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 d | lays) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 d | ays) |
| Б ( | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| Events All seizures | XXX | XXX | NA A AN A AN A | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 c | lays) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 d | ays) |
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 4 (0-3 o | lays) | | Dose 4 (4-7 | days) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0-3 | days) | | All Doses (4- | 7 days) | | All Doses (0-7 | days) |

| | | All Doses (0-3 | days) | | All Doses (4- | / days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at risk | Incidence Rate per 1000 person<br>days (95% CI) | Number of events<br>(n) | Person days at<br>risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) | Number of events (n) | Person days at risk<br>(n) | Incidence Rate per 1000 person<br>days (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Table 5.1.3 Incidence | e Rates (Per 1000 Per | rson Days) of Safety O | utcomes of Interest - Prospective Cohort Stu | dy (by Gender) | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Male | | | | |
| | | Dose 1 | (0-3 days) | | Dose | 1 (4-7 days) | | Dose 1 | 1 (0-7 days) |
| Events | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | 2 (0-3 days) | | Dose 2 | 2 (4-7 days) | | Dose 2 | 2 (0-7 days) |
| Events | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | 3 (0-3 days) | | Dose 3 | 3 (4-7 days) | | Dose 3 | 3 (0-7 days) |
| Events | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | 4 (0-3 days) | | Dose 4 | 4 (4-7 days) | | Dose 4 | 4 (0-7 days) |
| Events | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days (95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dos | es (0-3 days) | | All Dos | es (4-7 days) | All Doses (0-7 days) | | |
| F | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose | 1 (0-7 days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures XXX XXX XXX (XX.X - XX.X) XXX X | XX.X (XX.X - XX.X) | | | | | | | | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | xxx xxx | | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | 2 (0-3 days) | | Dose 2 | 2 (4-7 days) | Dose 2 (0-7 days) | | |
| Events | events | risk | Incidence Rate per 1,000 person days<br>(95%CI) | events | risk | | events | risk | Incidence Rate per 1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | 3 (0-3 days) | | Dose 3 | 3 (4-7 days) | | Dose 3 | 3 (0-7 days) |
| Events | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | 4 (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 | 4 (0-7 days) |
| Events | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dos | ses (0-3 days) | | All Dos | es (4-7 days) | | All Dos | ses (0-7 days) |
| Events | Number of events (n) | Person days at risk (n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events | Person days at risk (n) | Incidence Rate per 1,000 person days<br>(95%CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per 1,000 person days<br>(95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and | | | | | | | ***** | ***** | NN N ANN N NN N |
| | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| angioedema Apnea | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) |

| | | | | Perma | nent residents | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of<br>events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of<br>events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | 2 (0-3 days) | | Dose 2 | (4-7 days) | | Dose 2 | 2 (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Jrticaria and<br>ingioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | 4 (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 | (0-7 days) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dos | es (0-3 days) | | All Dose | es (4-7 days) | | All Dose | es (0-7 days) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| 2,010 | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |


| Urticaria and | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| angioedema | | | , | | | ` | ΛΛΛ | | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Tempo | rary residents | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 | (0-7 days) |
| | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| Events | | | | | | | | () | _ |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | 2 (0-3 days) | | Dose 2 | (4-7 days) | | Dose 2 | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 3 | (0-3 days) | | Dose 3 | (4-7 days) | Dose 3 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | (4-7 days) | | (0-7 days) | |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| | ****** | ***** | W. V. AW. V. W. V. | ***** | ***** | | ****** | ***** | ****************** |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | | All Dos | es (4-7 days) | | All Dos | es (0-7 days) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Table 5.1.5 Incidence Rates (Per 1000 Person Days) of Safety Outcomes of Interest - Prospective cohort study (by Co-administration of other vaccines on the same date)

| | | | Co-administrat | tion of other vacc | ines on the same o | late (Yes)* | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 d | lays) | Dose 1 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 d | lays) | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | xxx | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 d | lays) | | Dose 3 (0-7 d | ays) |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X(XX.X - XX.X) $XX.X(XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X<br>XX.X (XX.X - XX.X |
| 1 COLLE SCIZUICS | 71/1/1 | АЛЛ | AA.A(AA.A-AA.A) | 71/1/1 | 71/11 | AA.A(AA.A - AA.A) | 71/1/1 | AAA | 11.11 (11.11 - 11.11 |

| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 o | days) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0- | 3 days) | | All Doses (4-7 | days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

## Co-administration of other vaccines on the same date (No)

Dose 1 (0-3 days) Dose 1 (4-7 days) Dose 1 (0-7 days)

| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 d | lays) | | Dose 2 (0-7 d | ays) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 d | lays) | | Dose 3 (0-7 d | ays) |
| F. A | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events (n) | Person days at risk (n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Urticaria and

angioedema Apnea

Fever

XX.X (XX.X - XX.X)

XX.X (XX.X - XX.X)

XX.X (XX.X - XX.X)

| Dos | | | days) | | Dose 4 (4-7 d | lays) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events (n) | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | 3 days) | | All Doses (4-7 | days) | All Doses (0-7 days) | | | |
| | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1000<br>person days (95% CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) | Number of events | Person days at<br>risk<br>(n) | Incidence Rate per<br>1000 person days<br>(95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X |

XXX

XXX

XXX

XXX

XXX

XXX

XX.X (XX.X - XX.X)

XX.X (XX.X - XX.X)

XX.X(XX.X - XX.X)

XXX

XXX

XXX

XXX

XXX

XXX

XX.X (XX.X - XX.X)

XX.X (XX.X - XX.X)

XX.X(XX.X - XX.X)

XXX

XXX

XXX

XXX

XXX

XXX

<sup>\*</sup>Any dose of 13vPnC has been vaccinated on the same day as the other vaccines.

| | | | | | Winter | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | Dose 1 (0-7 days) | | |
| Events | Number of<br>events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of<br>events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of<br>events<br>(n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 | (4-7 days) | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 (0 | 0-7 days) |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | All Dos | es (4-7 days) | All Doses (0-7 days) | | | |
| Essente | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | | Spring | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 (0 | 0-7 days) |
| F4- | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 | (4-7 days) | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | 373737 | ****** | WWW | 373737 | **************************** | www | 3/3/3/ | VV V (VV V VV V) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 3 | (0-3 days) | | Dose 3 | (4-7 days) | | Dose 3 ( | )-7 days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | Dose 4 (4-7 days) | | | Dose 4 (0-7 days) | | |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0-3 days) | | | All Dos | es (4-7 days) | All Doses (0-7 days) | | |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |

| Number of events (n) XXX XXX XXX XXX | Person days at risk (n) XXX XXX XXX XXX XXX | (0-3 days) Incidence Rate per 1,000 person days (95%CI) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | Number of events (n) XXX XXX XXX XXX XXX | Dose 1 Person days at risk (n) XXX XXX XXX XXX XXX | (4-7 days) Incidence Rate per 1,000 person days (95%CI) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | Number of events (n) XXX XXX XXX XXX | Dose 1 (0 Person days at risk (n) XXX XXX XXX XXX XXX | Incidence Rate per 1,00 person days (95%CI) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|
| events<br>(n)<br>XXX | Person days<br>at risk<br>(n)<br>XXX | Incidence Rate per 1,000 person days (95%CI) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | Number of events (n) XXX XXX | Person days<br>at risk<br>(n)<br>XXX | Incidence Rate per 1,000 person days (95%CI) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | events (n) XXX XXX | Person<br>days at risk<br>(n)<br>XXX | Incidence Rate per 1,00<br>person days (95%CI) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) |
| events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of<br>events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | events<br>(n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,00<br>person days (95%CI)<br>XX.X (XX.X - XX.X) |
| events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of<br>events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | events<br>(n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,00<br>person days (95%CI) |
| events | Person days<br>at risk | Incidence Rate per 1,000 person | Number of events | Dose 1 Person days at risk | Incidence Rate per 1,000 person | events | Person<br>days at risk | Incidence Rate per 1,00 |
| | Dose 1 | (0-3 days) | | | (4-7 days) | | Dose 1 (0 | 1-7 days) |
| | | | | Summer | | | | |
| XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | XXX<br>XXX | xxx xxx xxx xxx xxx xxx xxx | XXX XXX XXX.X (XX.X - XX.X) XXX XXX XX.X (XX.X - XX.X) XXX XXX XX.X (XX.X - XX.X) | XXX XXX XXX (XX.X - XX.X) XXX XXX XXX XXX (XX.X - XX.X) XXX XXX XXX XXX (XX.X - XX.X) XXX | XXX XXX XXX (XX.X - XX.X) XXX XXX XXX XXX XXX (XX.X - XX.X) XXX XXX XXX XXX XXX (XX.X - XX.X) XXX XXX | XXX XXX XXX XXX XXX (XX.X - XX.X) XXX XXX XXX (XX.X - XX.X) XXX XXX XXX (XX.X - XX.X) XXX XXX XXX (XX.X - XX.X) XXX XXX XXX (XX.X - XX.X) | XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX <td>XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX XXX</td> | XXX XXX |

| Urticaria and | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | (0-3 days) | | Dose 3 | (4-7 days) | Dose 3 (0-7 days) | | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 (4-7 days) | | | Dose 4 (0-7 days) | |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dos | es (0-3 days) | | All Doses (4-7 days) | | | All Doses (0-7 days) | |

| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | | Fall | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 (0 | 0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 2 (0-3 days) | | | | Dose 2 | (4-7 days) | Dose 2 (0-7 days) | | |
| Events | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |

| Security Service Ser | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Angle Angl | All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Mumber of Person days Max Ma | Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Number of cevents | Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Number of events Person days Incidence Rate per 1,000 person days Incidence Rate per 1,0 | Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Number of events Person days at risk (n) Incidence Rate per 1,000 person days (systell) Number of events (n) Incidence Rate per 1,000 person days (95%CI) Number of events (n) Incidence Rate per 1,000 person days (95%CI) | Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Number of vents Number of Number of vents Number of vents Number of vents Number of Number of vents Number of vents Number of vents Number of Number of vents Number of vents Number of vents Number of Number of vents Number | | | Dose 3 | 3 (0-3 days) | | Dose 3 | (4-7 days) | | Dose 3 ( | 0-7 days) |
| Seizures | Events | events | at risk | | events | at risk | Incidence Rate per 1,000 person<br>days (95%CI) | events | days at risk | Incidence Rate per 1,000<br>person days (95%CI) |
| berile seizures | Zyenes | | | | | | | | | |
| | All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Number of events Number of events Number of events (n) | Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Number of events Number of events Number of events Incidence Rate per 1,000 person days (95%CI) Number of events (n) Number of event | Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Number of events (n) Incidence Rate per 1,000 person days (95%CI) Number of events (n) Number of (n) | Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Number of events (n) Incidence Rate per 1,000 person days (95%CI) Number of events (n) Incidence Rate | Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| events (n) at risk (n) days (95%CI) events (n) at risk (n) days (95%CI) events (n) days at risk (n) person days (95%CI) events (n) events (n) days (95%CI) events (n) even | | | Dose 4 | 4 (0-3 days) | | Dose 4 | (4-7 days) | Dose 4 (0-7 days) | | |
| ebrile seizures XXX X | Events | events | at risk | | events | at risk <sup>°</sup> | | events | days at risk | |
| ebrile seizures XXX XXX XXX XXXX XXXX XXX XXX XXX XXX | | | | | | | | | | |
| Irticaria and ngioedema XXX XXX XXX XXX XXXX XXX XXX XXX XXX | All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| ngioedema XXX XXX XX.X (XX.X - XX.X) XXX XXX XXX XXX XX.X (XX.X - XX.X) XXX XXX XXX (XX.X - XX.X) | Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| pnea XXX XXX XXX (XX.X - XX.X) XXX X | Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| | | All Dose | es (0-3 days) | | All Dos | es (4-7 days) | | All Doses | (0-7 days) |
| Events | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) | Number of events (n) | Person<br>days at risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 ( | 0-3 days) | | Dose 1 (4 | l-7 days) | | Dose 1 | (0-7 days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%Cl) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 2 (0-3 days) | | | | Dose 2 (4 | I-7 days) | | Dose 2 | (0-7 days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 3 (0-3 days) | | | | Dose 3 (4-7 days) | | | Dose 3 | (0-7 days) |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 ( | 0-3 days) | | Dose 4 ( | 4-7 days) | | | (0-7 days) |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses | (0-3 days) | | All Doses | (4-7 days) | | All Dose | es (0-7 days) |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| NIS Protocol | I <b1851193></b1851193> |
|--------------|-------------------------|

## Statistical Analysis Plan

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Table 5.2.2 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest - Prospective cohort study (Age Stratification)

| | | | | Age 0- ≤ | 2 months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | | Dose 1 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | ys) | | Dose 2 (0-7 | days) |
| F 4 | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | XXX | XXX | () | XXX | | XX.X (XX.X - XX.X) | | | |

| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4-7 d | lays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Age 2- ≤4 months

Dose 1 (0-3 days) Dose 1 (4-7 days) Dose 1 (0-7 days)

| P | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| Events All seizures | XXX | XXX | WWW WWW WWW | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) $XX.X(XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) |
| | AAA | AAA | XX.X (XX.X - XX.X) | AAA | AAA | AA.A (AA.A - AA.A) | AAA | AAA | AA.A (AA.A - AA.A) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | ys) | | Dose 2 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | 717171 | 212121 | XX.X (XX.X - XX.X) | 212121 | 717171 | (111.11 111.11) | 717171 | 212121 | (222.22 222.21) |

| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | | All Doses (0- | 7 days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 4- ≤ | 6 months | | | | |
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | | Dose 1 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | ys) | | Dose 2 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | Dose 3 (0-7 days) | | |
| Events | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 4 (0-3 days) | | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Age 6- ≤8 months | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Dose 2 (4-7 days)

Dose 2 (0-7 days)

Dose 2 (0-3 days)

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | VVV | | VVV | VVV | VV V (VV V VV V) | | VVV | VVV (VV V VVV) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0-3 days) | | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 8- ≤ | 10 months | | | | |
| | | Dose 1 (0- | 3 days) | | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
| T | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses<br>(n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | VVV (VV V VVV) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0- | 3 days) | | Dose 2 (4-7 da) | ys) | | Dose 2 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0- | 3 days) | | Dose 3 (4-7 da | ys) | Dose 3 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0- | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | | | | 3/3/3/ | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0 | 0-3 days) | | All Doses (4-7 d | lays) | | All Doses (0- | 7 days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| A 00 1 | 0 /12 | months |
|--------|----------|--------|
| Age I | U- < I Z | months |

| | | Dose 1 (0-3 days) | | | Dose 1 (4-7 days) | | | Dose 1 (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |

| | | Dose 2 (0-3 days) | | | Dose 2 (4-7 da | ys) | Dose 2 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Dose 3 (0-3 days) Dose 3 (4-7 days) Dose 3 (0-7 days)

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | | All Doses (0-7 | 7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 12-≤ | 14 months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | ys) | | Dose 2 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| | Dose 1 (0-3 days) | | | | Dose 1 (4-7 da | ys) | | Dose 1 (0-7 | days) |
| | | | | Age 14- ≤ | 16 months | | | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | | All Doses (0- | 7 days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| angioedema Apnea | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) |
| Febrile seizures Urticaria and | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of<br>events<br>(n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | Dose 4 (0-7 days) | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and | | | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ | | | ( | | | ( |
| angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0- | 3 days) | | Dose 2 (4-7 da | ys) | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0- | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| F4- | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 4 (0-3 days) | | | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |

| All seizures<br>Febrile seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0-3 days) | | | All Doses (4-7 d | lays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |

| | | Dose 1 (0-3 | days) | | Dose 1 (4-7 days) | | | Dose 1 (0-7 days) | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 da | vs) | | Dose 2 (0-7 | davs) |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 da | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | · | XXX | XXX | |
| Febrile seizures | λλλ | λλλ | XX.X (XX.X - XX.X) | λλλ | λλλ | XX.X (XX.X - XX.X) | λλλ | λλλ | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Age 18- ≤ | 20 months | | | | |
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
| T | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses<br>(n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) $XX.X (XX.X - XX.X)$ | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da) | ys) | | Dose 2 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | xxx | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 davs) | | Dose 3 (4-7 da | vs) | | Dose 3 (0-7 | davs) |
| | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | | | | | | | | |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | | 7/7/7/ | | 7777 | 3/3/3/ | ************************************** | NAM. | 77777 | WWW WWW WWW |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0 | -3 days) | | All Doses (4-7 d | ays) | | All Doses (0- | 7 days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Age 20- $\leq$ 22 months | Age | 20- | <22 | months |
|--------------------------|-----|-----|-----|--------|
|--------------------------|-----|-----|-----|--------|

| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 da | ys) | Dose 1 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 da | ys) | Dose 2 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Dose 3 (0-3 days) Dose 3 (4-7 days) Dose 3 (0-7 days)

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 (0 | 3 days) | | Dose 4 (4-7 da | ys) | | Dose 4 (0-7 | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0 | )-3 days) | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events | VVV | VVV | | VVV | VVV | VV V (VV V VV V) | VVV | VVV | VV V (VV V VV V) |
| All seizures Febrile seizures | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) | XXX<br>XXX | XXX<br>XXX | XX.X (XX.X - XX.X)<br>XX.X (XX.X - XX.X) |
| | ΛΛΛ | ΛΛΛ | XX.X (XX.X - XX.X) | ΛΛΛ | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ | ΛΛΛ | ΛΛΛ | $\Lambda\Lambda.\Lambda (\Lambda\Lambda.\Lambda - \Lambda\Lambda.\Lambda)$ |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Age 22- ≤ | 24 months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0- | 3 days) | | Dose 1 (4-7 da) | ys) | Dose 1 (0-7 days) | | |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0 | 3 days) | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses<br>(n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0- | 3 days) | | Dose 3 (4-7 da) | ys) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 da | ys) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0-3 days) | | | All Doses (4-7 d | ays) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 1 | (0-3 days) | Male Dose 1 (4-7 days) | | | Dose 1 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 2 (0-3 days) | | | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 4 (0-3 days) | | | Dose 4 (4-7 days) | | | Dose 4 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | All Doses (0-3 days) | | | All Doses (4-7 days) | | | All Doses (0-7 days) | | |
| | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
|---|---|---|---|---|---|---|---|---|---|--|--|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| | | | | Fem | ale | | | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 (4-7 days) | | | Dose 1 (0-7 days) | | | |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | | |
| Events | | | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| | Dose 2 (0-3 days) | | | Dose 2 (4-7 days) | | | Dose 2 (0-7 days) | | | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | | |
| | | Dose 3 | (0-3 days) | | Dose 3 (4-' | 7 days) | | Dose 3 | (0-7 days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of<br>events<br>(n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 (4-' | 7 days) | | Dose 4 | (0-7 days) |
| Events | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of<br>events<br>(n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | s (0-3 days) | | All Doses (4 | -7 days) | | All Dose | es (0-7 days) |
| Events | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | | | Perm | anent residents | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 ( | 0-3 days) | | Dose 1 (4 | 4-7 days) | | Dose 1 | (0-7 days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 ( | 0-3 days) | | Dose 2 (4 | 1-7 days) | | Dose 2 | (0-7 days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 4 (0-3 days) | | 0-3 days) | | Dose 4 (4 | 4-7 days) | | Dose 4 | (0-7 days) |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses | (0-3 days) | | All Doses | (4-7 days) | | All Dose | es (0-7 days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | Temp | orary residents | | | | |
| | | Dose 1 ( | 0-3 days) | | Dose 1 ( | 4-7 days) | | Dose 1 | (0-7 days) |
| Essente | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 ( | 0-3 days) | | Dose 2 ( | 4-7 days) | | Dose 2 | 2 (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 3 ( | 0-3 days) | | Dose 3 (4 | 1-7 days) | | Dose 3 | (0-7 days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 ( | 0-3 days) | | Dose 4 (4 | 1-7 days) | | Dose 4 | (0-7 days) |
| Events | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95%CI) | Number of events | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses | (0-3 days) | | All Doses | (4-7 days) | | All Dose | es (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95%CI) | Number of events (n) | Person<br>days at<br>risk<br>(n) | Incidence Rate per 1,000<br>person days (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

Table 5.2.5 Incidence Rates (Per 1000 Doses) of Safety Outcomes of Interest - Prospective cohort study (by Co-administration of other vaccines on the same date)

| | | | Co-administrati | ion of other vacci | nes on the same | date (Yes)* | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 (0-3 | 3 days) | | Dose 1 (4-7 | days) | | Dose 1 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | 3 days) | | Dose 2 (4-7 | days) | Dose 2 (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | 3 days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 | days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 4 (0-3 | 3 days) | | Dose 4 (4-7 | days) | Dose 4 (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | All Doses (0 | -3 days) | | All Doses (4- | 7 days) | All Doses (0-7 days) | | |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

## Co-adminstration of other vaccines on the same date (No)

Dose 1 (0-3 days) Dose 1 (4-7 days) Dose 1 (0-7 days)

| Events | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
|---|---|---|---|---|---|---|---|---|---|
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 (0-3 | days) | | Dose 2 (4-7 | days) | | Dose 2 (0-7 c | days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 (0-3 | days) | | Dose 3 (4-7 | days) | | Dose 3 (0-7 o | days) |
| _ | Number of events | Number of doses | Incidence Rate per 1,000<br>doses (95% CI) | Number of events | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) |
| Events All seizures | XXX | XXX | VV V (VV V VV V) | XXX | XXX | VV V (VV V VV V) | XXX | XXX | VV V (VV V VV V) |
| | | | XX.X (XX.X - XX.X) | | | XX.X (XX.X - XX.X) | | | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| | | Dose 4 (0-3 | days) | | Dose 4 (4-7 c | days) | | Dose 4 (0-7 | days) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses (0- | -3 days) | | All Doses (4-7 | ' days) | | All Doses (0-7 | 7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000<br>doses (95% CI) | Number of events (n) | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) | Number of events | Number of doses (n) | Incidence Rate per<br>1,000 doses (95% CI) |
| All seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

<sup>\*</sup>Any dose of 13vPnC has been vaccinated on the same day as the other vaccines.

| | | | (0.2.1) | | Winter | <b>4-</b> • • | | | (0 <b>-</b> 1 |
|---|---|---|---|---|---|---|---|---|---|
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 | (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of<br>events<br>(n) | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of<br>events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 perso<br>days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 | (4-7 days) | | Dose 2 | (0-7 days) |
| Events | Number of events (n) | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 perso<br>days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| 2,010 | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 | 4 (0-7 days) |
| | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Dose | s (0-3 days) | | All Dose | s (4-7 days) | | All Dos | es (0-7 days) |
| | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of<br>events<br>(n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 perso<br>days (95%CI) |
| | | Dose 2 | (0-3 days) | | Dose 2 | (4-7 days) | | Dose 2 | (0-7 days) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Events | (n) | (n) | (-2) | (n) | (n) | , | (n) | (n) | ,() |
| | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Person days<br>at risk | Incidence Rate per 1,000 perso<br>days (95%CI) |
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 | (0-7 days) |
| | | | | | Spring | | | | |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Urticaria and | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| angioedema | | | | | | , | | | |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | (0-3 days) | | Dose 3 | (4-7 days) | | Dose 3 | 6 (0-7 days) |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000 doses (95%CI) | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 | l (0-7 days) |
| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X(XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | AUD | s (0-3 days) | | | s (4-7 days) | | | es (0-7 days) |

| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | | Summer | | | | |
| | | Dose 1 | (0-3 days) | | | (4-7 days) | | Dose 1 | (0-7 days) |
| | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| Events | (11) | (11) | | (11) | (11) | | (11) | (11) | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 2 | (0-3 days) | | Dose 2 | (4-7 days) | | Dose 2 | 2 (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 3 | (0-3 days) | | Dose 3 | (4-7 days) | | Dose 3 | 3 (0-7 days) |
| | Number of events (n) | Number of doses | Incidence Rate per 1,000 doses (95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000 doses (95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 | 1 (0-7 days) |
| | Number of events | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | All Doses | s (0-3 days) | | All Doses | (4-7 days) | | All Dos | es (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | | | Fall | | | | |
| | | Dose 1 | (0-3 days) | | Dose 1 | (4-7 days) | | Dose 1 | (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and<br>angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |

| Events | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
|---|---|---|---|---|---|---|---|---|---|
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | Dose 3 (0-3 days) | | | | Dose 3 | (4-7 days) | | Dose 3 (0-7 days) | |
| | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| Events | | | | | | | | | |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | Dose 4 | (0-3 days) | | Dose 4 | (4-7 days) | | Dose 4 | 4 (0-7 days) |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |

| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Apnea | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Fever | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | All Doses (0-3 days) | | | All Doses (4-7 days) | | | All Doses (0-7 days) | | |
| Events | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Number of doses (n) | Incidence Rate per 1,000 doses<br>(95%CI) | Number of events (n) | Person days<br>at risk<br>(n) | Incidence Rate per 1,000 person<br>days (95%CI) |
| All Seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| Febrile seizures | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | ΛΛΛ | AA.A(AA.A-AA.A) | 2020 | 717171 | 717171 (71717171 717171) | | | ` ' |
| Urticaria and angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) |
| | | | ` ' | | | , | | | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) |
| angioedema | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | XX.X (XX.X - XX.X) | XXX | XXX | , |

Table~6.~Validation~of~ICD~code~using~adjudicated~safety~outcome~based~on~medical~records~of~children~as~gold~standard:~Positive~Predictive~Value~(PPV)

| | 25.4.6.1 | |
|---|---|---|
| Outcome | Main Study | Prospective Cohort Study |
| Seizures (including febrile seizures) | a/n1<br>PPV (%) | a/n1<br>PPV (%) |
| Urticaria and angioedema | a/n1<br>PPV (%) | a/n1<br>PPV (%) |
| Apnea | a/n1<br>PPV (%) | a/n1<br>PPV (%) |
| Fever | a/n1<br>PPV (%) | a/n1<br>PPV (%) |

Note: a= agreed outcome b/w cohort identified and adjudicated outcome n1=cohort identified outcome

## Table 6.1.1 Validation of ICD code (Main Study): Seizures (including febrile seizures)

| Main Study Results | Adjudication Results | |
|--------------------|----------------------|----|
| | Yes | No |
| Yes | | |
| No | | |

## Table 6.1.2 Validation of ICD code (Main Study): Urticaria and angioedema

| Main Study Results | Adjudicati | on Results |
|--------------------|------------|------------|
| | Yes | No |
| Yes | | |
| No | | |

| Table 6.1.3 Validation of ICD code (Main Study): Apnea | | | | |
|---|---|---|---|---|
| Main Study Results | Adj | udicatio | n Results | |
| | Yes | | No | |
| | 100 | | 110 | |
| Yes | | | | |
| No | | | | |
| Table 6.1.4 Validation of ICD code (Main Study) | : Fever | | | |
| Main Study Results | Adj | udicatio | n Results | |
| | V | | Ma | |
| | Yes | | No | |
| Yes | | | | |
| No | | | | |
| Table 6.2.1 Validation of ICD code (Prospective Seizures (including febrile seizures) | Study): | | | |
| Prospective Study Results | | | Adjudication | n Results |
| | | | X7 | N |
| | | | Yes | No |
| Yes | | | | |
| No | | | | |
| Table 6.2.2 Validation of ICD code (Prospective Study):<br>Urticaria and angioedema | | | | |
| Prospective Study Results | | | Adjudication | n Results |
| | | | 37 | 3.7 |
| | | | Yes | No |
| Yes | | | | |
| No | | | | |
| 110 | | <u> </u> | | |

| Table 6.2 3 Validation of ICD code (Prospective Study): Apnea | | | | | |
|---|---|---|---|---|---|
| Prospective cohort study Results | | Adjudication Results | | | |
| | | Y | es | No | |
| Yes | | | | | |
| No | | | | | |
| Table 6.2.4 Validation of ICD code (Prospective co | hort study): | Fever | | | |
| Prospective Study Results | | A | djudication | Results | |
| | | Y | es | No | |
| Yes | | | | | |
| No | | | | | |
| Table 7. Validation of ICD code using adjudicated reference standard: Sensitivity and Specificity | safety outco | | | | |
| Outcome Seizures (including febrile seizures) | | Sensitivi | ty | Specific | ity |
| Apnea | | | | | |
| | | <u> </u> | | | |
| Table 7.1.1 Validation of ICD code using adjudicated safety outcome in the Prospective Cohort Study as a reference standard: Seizures (including febrile seizures) | | | | | |
| | Adjudicated Prospective cohort study<br>Results | | | | |
| Main Study Results | Adjudicate | | ts | | |
| Main Study Results | Adjudicate<br>Ye. | Resul | ts<br>No | | |

| No |
|----|

Table 7.1.2 Validation of ICD code using adjudicated safety outcome in the Prospective Cohort Study as a reference standard: Apnea

| Main Study Results | Adjudicated Prospec | |
|--------------------|---------------------|----|
| | Yes | No |
| Yes | | |
| No | | |

Table 8. Validation of ICD code using the reported terms by parents/legal guardians in the Prospective Cohort Study as a non-reference standard: Positive Percentage Agreement (PPA) and Negative Percentage Agreement (NPA)

| Outcome | Positive Percentage Agreement<br>(PPA) | Negative Percentage Agreement (NPA) |
|---|---|---|
| Urticaria and angioedema | | |
| Fever | | |

Table 8.1.1 Validation of ICD code using the reported terms by parents/legal guardians in the Prospective Cohort Study as a non-reference standard: Urticaria and angioedema

| Main Study Results | Reported Prospecti<br>Resul | |
|--------------------|-----------------------------|----|
| | Yes | No |
| Yes | | |
| No | | |

Table~8.1.2~Validation~of~ICD~code~using~the~reported~terms~by~parents/legal~guardians~in~the~Prospective~Cohort~Study~as~a~non-reference~standard:~Fever

| Main Study Results | Reported Prospective cohort study<br>Results | |
|--------------------|----------------------------------------------|----|
| | Yes | No |
| Yes | | |
| No | | |

## **Document Approval Record**

**Document Name:** B1851193\_STATISTICAL ANALYSIS PLAN\_MAIN ANALYSIS\_CLEA

N\_07 JAN 2021

**Document Title:** B1851193\_STATISTICAL ANALYSIS PLAN\_MAIN ANALYSIS\_CLEA

N\_07 JAN 2021

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|-------------------|
| PPD | 08-Jan-2021 15:58:42 | Scientific Review |